CLINICAL TRIAL: NCT03234036
Title: A Two Part Study to Assess i) the Relative Bioavailability and Food Effect of a Novel Tablet Formulation of Boosted-GSK2838232 Compared to Capsule and ii) the Safety and Pharmacokinetics of Repeated Once-Daily Doses of Non-boosted GSK2838232
Brief Title: A Two-part Study to Compare a Tablet and Capsule Formulation of GSK2838232 With and Without Food, and to Assess the Safety and Drug Levels of Repeated Once-daily Doses of GSK2838232 Without Ritonavir
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: GlaxoSmithKline (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Crossover | Masking: Double | Purpose: Treatment
Other Study IDs: 205820
Record Dates: First submitted 2017-07-26; First posted 2017-07-31 (Actual); Results first posted 2019-03-07 (Actual); Last update posted 2020-10-28 (Actual); Status verified 2020-10

CONDITIONS: Infection, Human Immunodeficiency Virus; HIV Infections
Keywords: GSK2838232; safety; food effect; capsule; healthy; PK; tablet
MeSH Terms: conditions — Infections; Acquired Immunodeficiency Syndrome; HIV Infections | interventions — GSK-2838232; Tablets; Ritonavir

STUDY DESIGN:
Intervention Model Description: The randomization number will determine the allocation of treatment sequences (ABC or BAC) for Part 1, and of treatment (GSK2838232 without RTV or placebo) for Part 2. Allocation to treatment for Part 1A or Part 1B (with Part 2 being fixed) will be according to a predetermined random order.
Who Masked: Participant, Investigator
Masking Description: Part 1 of the study will be open label and thus not be blinded. Part 2 of the study will be single blinded because of the unavailability of matching placebo tablets. The Principal Investigator and the subject will be completely blinded to specific treatment assignment.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (4):
- Treatment sequence ABC: Part 1 (Experimental): A single dose of GSK2838232 200 mg (as 4 x 50 mg) capsule formulation will be administered under fed conditions (treatment A) in period 1 in Part 1A.
  A single dose of GSK2838232 200 mg (as 2 x 100 mg) tablet formulation will be administered under fed conditions (treatment B) in period 2 in Part 1A.
  Both these treatments in Part 1A will be administered with RTV in fed state with a washout of 10 days.
  A single dose of GSK2838232 200 mg (as 2 x 100 mg) tablet formulation (with RTV) will be administered under fasted conditions (treatment C) in period 3 in Part 1B.
  There will be a wash out of 15 days between Part 1A and Part 1B.
  Interventions: Drug: GSK2838232 100 mg tablet; Drug: GSK2838232 50 mg capsule; Drug: Ritonavir 100 mg tablets
- Treatment sequence BAC: Part 1 (Experimental): A single dose of GSK2838232 200 mg (as 2 x 100 mg) tablet formulation will be administered under fed conditions (treatment B) in period 1 in Part 1A.
  A single dose of GSK2838232 200 mg (as 4 x 50 mg) capsule formulation will be administered under fed conditions (treatment A) in period 2 in Part 1A.
  A single dose of GSK2838232 200 mg (as 2 x 100 mg) tablet formulation (with RTV) will be administered under fasted conditions (treatment C) in period 3 in Part 1B.
  There will be a wash out of 15 days between Part 1A and Part 1B.
  Interventions: Drug: GSK2838232 100 mg tablet; Drug: GSK2838232 50 mg capsule; Drug: Ritonavir 100 mg tablets
- GSK2838232 tablet without RTV: Part 2 (Experimental): In Part 2, subjects will receive non-RTV boosted GSK2838232 500 mg, given as single daily doses for 11 days. The dose will not exceed 500 mg (as 5 x 100 mg tablets) once daily (QD).
  Interventions: Drug: GSK2838232 100 mg tablet
- Placebo without RTV: Part 2 (Placebo Comparator): In Part 2, subjects will receive a Placebo given as single daily doses for 11 days.
  Interventions: Drug: Placebo for GSK2838232 tablets

INTERVENTIONS:
Drug: GSK2838232 100 mg tablet — It is a white to slightly colored tablet. It will be supplied as prefilled tablets in bulk for dispensing to subjects at the site according to the treatment code.
  Arms: GSK2838232 tablet without RTV: Part 2; Treatment sequence ABC: Part 1; Treatment sequence BAC: Part 1
Drug: GSK2838232 50 mg capsule — It is a pink unmarked capsule. It will be supplied as prefilled capsules in bulk for dispensing to subjects at the site according to the treatment code.
  Arms: Treatment sequence ABC: Part 1; Treatment sequence BAC: Part 1
Drug: Ritonavir 100 mg tablets — It is a white film-coated ovaloid tablets.
  Arms: Treatment sequence ABC: Part 1; Treatment sequence BAC: Part 1
Drug: Placebo for GSK2838232 tablets — It is a white to slightly colored tablet. The placebo tablets supplied will not be identical to GSK2838232 tablets. It will be administered by site staff via an opaque card or paper tube.
  Arms: Placebo without RTV: Part 2

SUMMARY:
This study will be conducted in two Parts to confirm the acceptability/selection of a tablet formulation for future clinical development of GSK2838232. Part 1 of the study will assess single ritonavir (RTV)-boosted doses of a new tablet formulation given with food (containing approximately 30% fat) against the reference capsule formulation also given with food and then will assess the impact of fasted conditions on the tablet performance. In Part 2, non-boosted GSK2838232 will be given as once-daily tablet doses for 11 days in a separate group of subjects, assuming the tablet performance is considered acceptable from Part 1. Approximately 16 healthy subjects will be enrolled to provide at least 12 evaluable subjects through the three study periods in Part 1. 10 healthy subjects will be enrolled to provide at least 8 evaluable subjects through the single study period in Part 2. The maximum duration of study participation will be approximately 9 to 10 weeks for Part 1; and 8 to 9 weeks for Part 2.

ELIGIBILITY:
Inclusion Criteria:

* Between 18 and 55 years of age inclusive, at the time of signing the informed consent.
* Healthy as determined by the Investigator or medically qualified designee based on a medical evaluation including medical history, physical examination, laboratory tests and cardiac monitoring.
* A subject with a clinical abnormality or laboratory parameter(s) which is/are not specifically listed in the inclusion or exclusion criteria, and outside the reference range for the population being studied, may be included only if the Investigator in consultation with the medical monitor, if required, agree and document that the finding is unlikely to introduce additional risk factors and will not interfere with the study procedures.
* A creatinine clearance (CLcr) > 80 milliliter per minute (mL/min) as determined by Cockcroft-Gault equation: CLcr = (140 minus age) multiplied by weight divided by (72 multiplied by serum creatinine) (times 0.85 if female) where age is in years, weight in kilogram (kg), and serum creatinine is in units of milligram per deciliter (mg/dL).
* Body weight >=50.0 kg (110 pounds [lbs.]) for men and >=45.0 kg (99 lbs) for women and body mass index (BMI) within the range 18.5 to 31.0 kg/meter (m)^2 (inclusive).
* Males or females.
* A female subject is eligible to participate if she is not pregnant (as confirmed by a negative serum human chorionic gonadotrophin [hCG] test), not lactating, and of non-reproductive potential which is defined as:

Reproductive potential:

There is no definitive drug-drug interaction (DDI) information with GSK2838232 and an interaction with oral contraceptives is possible, so other (barrier, inter-uterine device etc.) methods of contraception will be required. Females of reproductive potential may only be enrolled if they are using two forms of complementary contraception, which must include at least one barrier method. They will be counseled on safer sex practices. Fertile females, who have an established, long-term lifestyle of sexual abstinence, or only same sex partners, require no other means of birth control.

Non-reproductive potential:

* Pre-menopausal females with one of the following: Documented tubal ligation; documented hysteroscopic tubal occlusion procedure with follow-up confirmation of bilateral tubal occlusion; hysterectomy; documented Bilateral Oophorectomy.
* Postmenopausal defined as 12 months of spontaneous amenorrhea in questionable cases a blood sample with simultaneous follicle stimulating hormone (FSH) and estradiol levels consistent with menopause. Females on hormone replacement therapy (HRT) must discontinue HRT to allow confirmation of post-menopausal status prior to study enrolment.

  * Male subjects with female partners of child bearing potential must comply with the following contraception requirements from the time of first dose of study medication until one week after the last dose of study medication.
* Vasectomy with documentation of azoospermia.
* Male condom plus partner use of one of the contraceptive options below: Contraceptive subdermal implant with a <1 percent rate of failure per year; intrauterine device or intrauterine system with a <1 percent rate of failure per year; oral contraceptive, either combined or progestogen alone or injectable progestogen; contraceptive vaginal ring; percutaneous contraceptive patches.

  * Capable of giving signed informed consent.

Exclusion Criteria:

* ALT >1.5 times upper limit of normal (ULN)
* Bilirubin >1.5 times ULN (isolated bilirubin >1.5 times ULN is acceptable if bilirubin is fractionated and direct bilirubin <35 percent).
* Current or chronic history of liver disease, or known hepatic or biliary abnormalities.
* Subjects who have asthma or a history of asthma.
* Medical history of cardiac arrhythmias or cardiac disease or a family or personal history of long QT syndrome.
* Unable to refrain from the use of prescription or non-prescription drugs, including vitamins, herbal and dietary supplements (including St John's Wort) within 7 days (or 14 days if the drug is a potential enzyme inducer) or 5 half-lives (whichever is longer) prior to the first dose of study medication, unless in the opinion of the Investigator and GlaxoSmithKline medical monitor, the medication will not interfere with the study procedures or compromise participant safety.
* History of regular alcohol consumption (within 6 months prior to screening or unable to refrain from alcohol use from 5 days prior to admission through the last blood sample collected) defined as:

  • For United States sites: an average weekly intake of >14 drinks for males or >7 drinks for females. One drink is equivalent to 12 gram of alcohol: 12 ounces (360 mL) of beer, 5 ounces (150 mL) of wine or 1.5 ounces (45 mL) of 80 proof distilled spirits.
* Regular use of tobacco- or nicotine- containing products within 6 months prior to screening. Unable to refrain from smoking from the Screening Visit through the last blood sample collected. As confirmed by a urine cotinine test.
* History of sensitivity to any of the study medications, or components thereof or a history of drug or other allergy that, in the opinion of the investigator or medical monitor, contraindicates their participation.
* Presence of hepatitis B surface antigen (HBsAg), or positive hepatitis C virus (HCV) test result at screening or within 3 months prior to first dose of study treatment.
* Screening or Baseline cardiac troponin I greater than the 99 percent cutoff (>0.045 nanogram [ng]/mL by the Dimension Vista cTnI assay) for a given assay.
* A positive pre-study drug/alcohol screen.
* A positive test for human immunodeficiency virus (HIV) antibody.
* Where participation in the study would result in donation of blood or blood products in excess of 500 mL within 56 days.
* The subject has participated in a clinical trial and has received an investigational product within the following time period prior to the first dosing day in the current study: 30 days, 5 half-lives or twice the duration of the biological effect of the investigational product (whichever is longer).
* Exposure to more than four new chemical entities within 12 months prior to the first dosing day.
* Exclusion Criteria for 24-hour Screening Holter:

  * Any symptomatic arrhythmia (except isolated extra systoles).
  * Sustained cardiac arrhythmias (such as atrial fibrillation or flutter, supraventricular tachycardia (>= 10 consecutive beats), complete heart block).
  * Non-sustained or sustained ventricular tachycardia (defined as >=3 consecutive ventricular ectopic beats).
  * Any conduction abnormality (including but not specific to left or right incomplete or complete bundle branch block, atrioventricular (AV) block [2nd degree or higher], Wolff Parkinson White (WPW) syndrome etc.).
  * Sinus Pauses >3 seconds.
  * 300 or more supraventricular ectopic beats in 24 hours.
  * 250 or more ventricular ectopic beats in 24 hours.
* Any clinically significant abnormal echocardiogram finding.
* Exclusion criteria for screening ECG (a single repeat is allowed for eligibility determination):

  * Heart rate <45 or >100 beats per minute (bpm) for males; <50 or >100 bpm for females
  * PR interval <120 or >220 milliseconds (msec)
  * QRS duration <70 or >120 msec
  * QTc interval (Fridericia's) >450 msec
  * Evidence of previous myocardial infarction (does not include ST segment changes associated with re-polarization).
  * Any conduction abnormality (including but not specific to left or right complete bundle branch block, AV block [2nd degree or higher], WPW syndrome).
  * Sinus Pauses >3 seconds.
  * Any significant arrhythmia which, in the opinion of the Investigator or GSK medical monitor, will interfere with the safety for the individual subject.
  * Non-sustained or sustained ventricular tachycardia (>=3 consecutive ventricular ectopic beats).

Ages: 18 Years to 55 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 26 (Actual)
Dates: Start 2017-08-02 (Actual); Primary Completion 2017-11-10 (Actual); Study Completion 2017-11-10 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: GSK Clinical Trials, Study Director — GlaxoSmithKline
Locations (1):
- GSK Investigational Site, Baltimore, Maryland, United States

IPD SHARING:
Plan to Share IPD: Yes
IPD for this study is available via the Clinical Study Data Request site.
Supporting Information: Study Protocol, SAP, ICF, CSR
Time Frame: IPD is available via the Clinical Study Data Request site (copy the URL below to your browser)
Access Criteria: Access is provided after a research proposal is submitted and has received approval from the Independent Review Panel and after a Data Sharing Agreement is in place. Access is provided for an initial period of 12 months but an extension can be granted, when justified, for up to another 12 months.
URL: https://www.clinicalstudydatarequest.com/Posting.aspx?ID=20589

REFERENCES:
- [Background] Johnson M, Jewell RC, Gan J, Dumont E, Burns O, Johns BA. A Phase 1 Study to Assess the Relative Bioavailability, Food Effect, and Safety of a Tablet Formulation of GSK2838232, a Novel HIV Maturation Inhibitor in Healthy Participants After Single and Repeated Doses. Clin Pharmacol Drug Dev. 2020 Nov;9(8):972-977. doi: 10.1002/cpdd.820. Epub 2020 Jun 18. PMID 32558338

RESULTS

PARTICIPANT FLOW:
Recruitment Details: This two-part study assessed the relative bioavailability and food effect of a novel tablet formulation of boosted-GSK2838232 compared to capsule along with safety and pharmacokinetics of repeated once-daily doses of non-boosted GSK2838232. This study was conducted at a single center in the United States.
Pre-assignment Details: Participants received GSK2838232 200 milligrams (mg)/ritonavir as capsule or tablet formulation in Part 1 and GSK2838232 500 mg or placebo in Part 2. A total number of 16 participants were enrolled in Part 1 of the study and 10 participants were enrolled in Part 2. In total, 26 participants were enrolled in the study.
Groups:
- GSK2838232 Capsule Fed/Tablet Fed/Tablet Fasted With Ritonavir: Eligible participants received a single dose of GSK2838232 200 mg (as 4 x 50 mg) capsule administered under fed conditions in treatment period 1 along with ritonavir 100 mg tablet to be taken with water in fed condition, followed by a single dose of GSK2838232 200 mg (as 2 x 10 mg) tablet administered under fed conditions in treatment period 2 along with ritonavir 100 mg tablet to be taken with water in fed condition, followed by a single dose of GSK2838232 200 mg (as 2 x 10 mg) tablet administered under fasted conditions in treatment period 3 along with ritonavir 100 mg tablet to be taken with water in fasted condition. Treatment period 1 and 2 were separated by a wash-out period of 10 days. Treatment period 2 and 3 were separated by 15 days wash-out period.
- GSK2838232 Tablet Fed/Capsule Fed/Tablet Fasted With Ritonavir: Eligible participants received a single dose of GSK2838232 200 mg (as 2 x 10 mg) tablet administered under fed conditions in treatment period 1 along with ritonavir 100 mg tablet to be taken with water in fed condition, followed by a single dose of GSK2838232 200 mg (as 4 x 50 mg) capsule administered under fed conditions in treatment period 2 along with ritonavir 100 mg tablet to be taken with water in fed condition, followed by a single dose of GSK2838232 200 mg (as 2 x 10 mg) tablet administered under fasted conditions in treatment period 3 along with ritonavir 100 mg tablet to be taken with water in fasted condition. Treatment period 1 and 2 were separated by a wash-out period of 10 days. Treatment period 2 and 3 were separated by 15 days wash-out period.
- Part 2: Placebo: Eligible participants received single daily doses of placebo tablet orally along with water in fed condition for 11 days.
- Part 2: GSK2838232 500 mg Tablet Fed: Eligible participants received non-ritonavir boosted GSK2838232 500 mg, given as single daily doses in fed condition for 11 days.
Period: Part 1: Treatment Period 1(Up to 7 Days)
Arm/Group | GSK2838232 Capsule Fed/Tablet Fed/Tablet Fasted With Ritonavir | GSK2838232 Tablet Fed/Capsule Fed/Tablet Fasted With Ritonavir | Part 2: Placebo | Part 2: GSK2838232 500 mg Tablet Fed
Started | 8 | 8 | 0 | 0
Completed | 8 | 8 | 0 | 0
Not Completed | 0 | 0 | 0 | 0
Period: Part 1:Washout Period 1 (Up to 10 Days)
Arm/Group | GSK2838232 Capsule Fed/Tablet Fed/Tablet Fasted With Ritonavir | GSK2838232 Tablet Fed/Capsule Fed/Tablet Fasted With Ritonavir | Part 2: Placebo | Part 2: GSK2838232 500 mg Tablet Fed
Started | 8 | 8 | 0 | 0
Completed | 7 | 7 | 0 | 0
Not Completed | 1 | 1 | 0 | 0
Not completed — Adverse Event | 1 | 1 | 0 | 0
Period: Part 1: Treatment Period 2(Up to 7 Days)
Arm/Group | GSK2838232 Capsule Fed/Tablet Fed/Tablet Fasted With Ritonavir | GSK2838232 Tablet Fed/Capsule Fed/Tablet Fasted With Ritonavir | Part 2: Placebo | Part 2: GSK2838232 500 mg Tablet Fed
Started | 7 | 7 | 0 | 0
Completed | 7 | 7 | 0 | 0
Not Completed | 0 | 0 | 0 | 0
Period: Part 1:Washout Period 2 (Up to 15 Days)
Arm/Group | GSK2838232 Capsule Fed/Tablet Fed/Tablet Fasted With Ritonavir | GSK2838232 Tablet Fed/Capsule Fed/Tablet Fasted With Ritonavir | Part 2: Placebo | Part 2: GSK2838232 500 mg Tablet Fed
Started | 7 | 7 | 0 | 0
Completed | 7 | 7 | 0 | 0
Not Completed | 0 | 0 | 0 | 0
Period: Part 1:Treatment Period 3 (Up to 7 Days)
Arm/Group | GSK2838232 Capsule Fed/Tablet Fed/Tablet Fasted With Ritonavir | GSK2838232 Tablet Fed/Capsule Fed/Tablet Fasted With Ritonavir | Part 2: Placebo | Part 2: GSK2838232 500 mg Tablet Fed
Started | 7 | 7 | 0 | 0
Completed | 7 | 7 | 0 | 0
Not Completed | 0 | 0 | 0 | 0
Period: Part 2 (Up to 25 Days)
Arm/Group | GSK2838232 Capsule Fed/Tablet Fed/Tablet Fasted With Ritonavir | GSK2838232 Tablet Fed/Capsule Fed/Tablet Fasted With Ritonavir | Part 2: Placebo | Part 2: GSK2838232 500 mg Tablet Fed
Started | 0 | 0 | 3 | 7
Completed | 0 | 0 | 3 | 7
Not Completed | 0 | 0 | 0 | 0

BASELINE CHARACTERISTICS:
Groups:
- Part 1: All Participants Receiving GSK2838232/Ritonavir: Eligible participants were assigned to treatment sequence AB or BA where A=single dose of GSK2838232 200 mg (as 4 x 50 mg) capsule under fed condition and B=single dose of GSK2838232 200 mg (as 4 x 50 mg) tablet formulations administered under fed condition in treatment periods 1 and 2 along with ritonavir 100 mg to be taken with water in fed condition. Participants received a single dose of GSK2838232 200 mg (as 2 x 10 mg) tablet administered under fasted conditions in treatment period 3 along with ritonavir 100 mg to be taken with water in fasted condition. Treatment periods 1 and 2 were separated by a wash-out period of 10 days. Treatment periods 2 and 3 were separated by a wash-out period of 15 days.
- Total: Total of all reporting groups
Arm/Group | Part 1: All Participants Receiving GSK2838232/Ritonavir | Part 2: Placebo | Part 2: GSK2838232 500 mg Tablet Fed | Total
Number analyzed (Participants) | 16 | 3 | 7 | 26
Age, Continuous [Mean (Standard Deviation); unit: Years] | 36.3 (9.54) | 41.0 (9.64) | 34.6 (7.81) | 36.38 (9.30)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 9 | 0 | 1 | 10
  Male | 7 | 3 | 6 | 16
Race/Ethnicity, Customized [Count of Participants; unit: Participants]
  BLACK OR AFRICAN AMERICAN | 8 | 2 | 6 | 16
  WHITE - WHITE/CAUCASIAN/EUROPEAN HERITAGE | 6 | 1 | 0 | 7
  MULTIPLE-ASIAN & BLACK OR AFRICAN AMERICAN | 2 | 0 | 0 | 2
  AMERICAN INDIAN OR ALASKA NATIVE | 0 | 0 | 1 | 1

OUTCOME MEASURES:

1. Primary Outcome: Part 1: Area Under the Concentration-time Curve From Time Zero (Pre-dose) Extrapolated to Infinite Time (AUC [0-infinity]) Following Administration of GSK2838232 Tablet and Capsule Formulation in Fed State
Description: Blood samples were collected at indicated time points for pharmacokinetic analysis of GSK2838232 given as tablet and capsule formulation in fed state. Pharmacokinetic parameters were determined using standard non-compartmental methods. Pharmacokinetic Population comprised of all participants in the Safety Population who had at least 1 non-missing pharmacokinetic assessment (Non-quantifiable [NQ] values were considered as non-missing values).
Time Frame: Pre-dose, 0.5, 1, 1.5, 2, 2.5, 3, 3.5, 4, 6, 8, 12, 24, 36, 48, 72, 96, and 120 hours post-dose in treatment periods 1 and 2 of Part 1
Population: Pharmacokinetic Population
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: Hours*nanogram per milliliter
Groups:
- Part 1: GSK2838232 200 mg/Ritonavir Capsule Fed: Participants received a single dose of GSK2838232 200 mg (as 4 x 50 mg) capsule formulation along with ritonavir 100 mg tablet administered under fed conditions in treatment periods 1 and 2.
- Part 1: GSK2838232 200 mg/Ritonavir Tablet Fed: Participants received a single dose of GSK2838232 200 mg (as 2 x 10 mg) tablet formulation along with ritonavir 100 mg tablet administered under fed conditions in treatment periods 1 and 2.
Arm/Group | Part 1: GSK2838232 200 mg/Ritonavir Capsule Fed | Part 1: GSK2838232 200 mg/Ritonavir Tablet Fed
Number analyzed (Participants) | 15 | 15
Hours*nanogram per milliliter | 4672.28 (40.68) | 4437.98 (30.83)

2. Primary Outcome: Part 1: Maximum Observed Concentration (Cmax) Following Administration of GSK2838232 Tablet and Capsule Formulation in Fed State
Description: Blood samples were collected at indicated time points for pharmacokinetic analysis of GSK2838232 given as tablet and capsule formulation in fed state. Pharmacokinetic parameters were determined using standard non-compartmental methods.
Time Frame: as for outcome 1
Population: Pharmacokinetic Population
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: Nanograms per milliliter
Arm/Group | Part 1: GSK2838232 200 mg/Ritonavir Capsule Fed | Part 1: GSK2838232 200 mg/Ritonavir Tablet Fed
Number analyzed (Participants) | 15 | 15
Nanograms per milliliter | 109.054 (48.01) | 118.118 (27.59)

3. Primary Outcome: Part 1: AUC (0-infinity) Following Administration of GSK2838232 Tablet in Fasted and Fed State
Description: Blood samples were collected at indicated time points for pharmacokinetic analysis of GSK2838232 given as tablet formulation in fed and fasted state. Pharmacokinetic parameters were determined using standard non-compartmental methods.
Time Frame: Pre-dose, 0.5, 1, 1.5, 2, 2.5, 3, 3.5, 4, 6, 8, 12, 24, 36, 48, 72, 96, and 120 hours post-dose in treatment periods 1, 2 and 3 of Part 1
Population: Pharmacokinetic Population
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: Hours*nanogram per milliliter
Groups:
- Part 1: GSK2838232 200 mg/Ritonavir Tablet Fed: Participants received a single dose of GSK2838232 200 mg (as 2 x 10 mg) tablet formulation administered under fed conditions in treatment periods 1 and 2 along with ritonavir 100 mg tablet to be taken with water in fed condition.
- Part 1: GSK2838232 200 mg/Ritonavir Tablet Fasted: Participants received a single dose of GSK2838232 200 mg (as 2 x 100 mg) tablet formulation under fasted conditions in treatment period 3 along with ritonavir 100 mg tablet to be taken with water in fasted condition.
Arm/Group | Part 1: GSK2838232 200 mg/Ritonavir Tablet Fed | Part 1: GSK2838232 200 mg/Ritonavir Tablet Fasted
Number analyzed (Participants) | 15 | 14
Hours*nanogram per milliliter | 4437.98 (30.83) | 1816.27 (36.42)

4. Primary Outcome: Part 1: Cmax Following Administration of GSK2838232 Tablet in Fasted and Fed State
Description: as for outcome 3
Time Frame: as for outcome 3
Population: Pharmacokinetic Population
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: Nanograms per milliliter
Arm/Group | Part 1: GSK2838232 200 mg/Ritonavir Tablet Fed | Part 1: GSK2838232 200 mg/Ritonavir Tablet Fasted
Number analyzed (Participants) | 15 | 14
Nanograms per milliliter | 118.118 (27.59) | 50.437 (35.61)

5. Primary Outcome: Part 1: Time of Occurrence of Cmax (Tmax) Following Administration of GSK2838232 Tablet in Fasted and Fed State
Description: as for outcome 3
Time Frame: as for outcome 3
Population: Pharmacokinetic Population
Measure: Median (Full Range); unit: Hours
Arm/Group | Part 1: GSK2838232 200 mg/Ritonavir Tablet Fed | Part 1: GSK2838232 200 mg/Ritonavir Tablet Fasted
Number analyzed (Participants) | 15 | 14
Hours | 5.983 [2.00 to 24.03] | 3.508 [2.00 to 11.97]

6. Primary Outcome: Part 2: Number of Participants With Serious Adverse Events (SAEs) and Non-SAEs
Description: An adverse event (AE) is any untoward medical occurrence in a clinical study participant, temporally associated with the use of a study treatment, whether or not considered related to the study treatment. SAE is defined as any untoward medical occurrence that, at any dose results in death, is life threatening, requires hospitalization or prolongation of existing hospitalization, results in persistent disability/incapacity, is a congenital anomaly/ birth defect, is associated with liver injury or impaired liver function or any other situations as per medical or scientific judgment. Safety Population comprised of all participants who received at least 1 dose of the study treatment (including placebo) with at least 1 post-Baseline safety assessment. Number of participants with SAEs and common non-SAEs (>=5%) are presented.
Time Frame: Up to 25 days
Population: Safety Population
Measure: Count of Participants; unit: Participants
Arm/Group | Part 2: Placebo | Part 2: GSK2838232 500 mg Tablet Fed
Number analyzed (Participants) | 3 | 7
Participants
  Any SAE | 0 | 0
  Any non-SAE | 1 | 0

7. Primary Outcome: Part 2: Number of Participants With Worst Case Hematology Results to Potential Clinical Importance (PCI) Criteria
Description: Blood samples were collected from participants for analysis of following hematology parameters; hematocrit, hemoglobin, leukocytes, lymphocytes, neutrophils and platelets. PCI ranges were < 0.075 or >0.54 proportion of red blood cells in blood for hematocrit, <25 or >180 grams per liter (g/L) for hemoglobin, < 3 or >20 cells per liter (cells/L) for leukocytes, 0.8 x10^9 cells/L for lymphocytes, 1.5 x10^9 cells/L for neutrophils, and <100 or >550 cells/L for platelets. Participants were counted in the worst case category that their value changes to (low, within range or no change, or high), unless there is no change in their category. Participants whose laboratory value category was unchanged (example given [e.g.], High to High), or whose value became within range, were recorded in the "To within Range or No Change" category.
Time Frame: Up to 25 days
Population: Safety Population
Measure: Count of Participants; unit: Participants
Arm/Group | Part 2: Placebo | Part 2: GSK2838232 500 mg Tablet Fed
Number analyzed (Participants) | 3 | 7
Participants
  Hematocrit; To Low | 0 | 0
  Hematocrit; To within Range or No Change | 3 | 7
  Hematocrit; To High | 0 | 0
  Hemoglobin; To Low | 0 | 0
  Hemoglobin; To within Range or No Change | 3 | 7
  Hemoglobin; To High | 0 | 0
  Leukocytes; To Low | 0 | 0
  Leukocytes; To within Range or No Change | 3 | 7
  Leukocytes; To High | 0 | 0
  Lymphocytes; To Low | 0 | 0
  Lymphocytes; To within Range or No Change | 3 | 7
  Lymphocytes; To High | 0 | 0
  Neutrophils; To Low | 1 | 1
  Neutrophils; To within Range or No Change | 2 | 6
  Neutrophils; To High | 0 | 0
  Platelets; To Low | 0 | 0
  Platelets; To within Range or No Change | 3 | 7
  Platelets; To High | 0 | 0

8. Primary Outcome: Part 2: Number of Participants With Worst Case Clinical Chemistry Results to PCI Criteria
Description: Blood samples were collected from participants for analysis of following clinical chemistry parameters; glucose, alanine aminotransferase (ALT), albumin, alkaline phosphatase, aspartate aminotransferase (AST), bilirubin, calcium, potassium and sodium. PCI ranges were <30 g/L for albumin, <2 or >2.75 millimoles per liter (mmol/L) for calcium, <3 or >9 mmol/L for glucose, >=2 times Upper limit of Normal (ULN) units per liter (U/L) for ALT, >=2 times ULN U/L for alkaline phosphatase, >=2 times ULN U/L for AST, >=1.5 times ULN micromoles per liter (µmol/L) for bilirubin, <3 or >5.5 mmol/L for potassium, and <130 or >150 mmol/L for sodium. Participants were counted in the worst case category that their value changes to (low, within range or no change,or high), unless there is no change in their category. Participants whose laboratory value category was unchanged (e.g., High to High), or whose value became within range, were recorded in the "To within Range or No Change" category.
Time Frame: Up to 25 days
Population: Safety Population
Measure: Count of Participants; unit: Participants
Arm/Group | Part 2: Placebo | Part 2: GSK2838232 500 mg Tablet Fed
Number analyzed (Participants) | 3 | 7
Participants
  Glucose; To Low | 0 | 0
  Glucose; To within Range or No Change | 3 | 7
  Glucose; To High | 0 | 0
  ALT; To Low | 0 | 0
  ALT; To within Range or No Change | 3 | 7
  ALT; To High | 0 | 0
  Albumin; To Low | 0 | 0
  Albumin; To within Range or No Change | 3 | 7
  Albumin; To High | 0 | 0
  Alkaline phosphatase; To Low | 0 | 0
  Alkaline phosphatase; To within Range or No Change | 3 | 7
  Alkaline phosphatase; To High | 0 | 0
  AST; To Low | 0 | 0
  AST; To within Range or No Change | 3 | 7
  AST; To High | 0 | 0
  Bilirubin; To Low | 0 | 0
  Bilirubin; To within Range or No Change | 3 | 7
  Bilirubin; To High | 0 | 0
  Calcium; To Low | 0 | 0
  Calcium; To within Range or No Change | 3 | 7
  Calcium; To High | 0 | 0
  Potassium; To Low | 0 | 0
  Potassium; To within Range or No Change | 3 | 7
  Potassium; To High | 0 | 0
  Sodium; To Low | 0 | 0
  Sodium; To within Range or No Change | 3 | 7
  Sodium; To High | 0 | 0

9. Primary Outcome: Part 2: Number of Participants With Worst Case Urinalysis Results Relative to Normal Range Criteria
Description: Urine samples were collected from participants for analysis of following urinalysis parameters; specific gravity, potential of hydrogen (pH), presence of glucose, protein, occult blood, ketones in urine analyzed by dipstick method. The dipstick test gives results in a semi-quantitative manner. Urine specific gravity is a measure of the concentration of solutes in the urine and provides information on the kidney's ability to concentrate urine. The reference range is 1.002-1.030. Urine pH is an acid-base measurement. Normal urine has a slightly acid pH (5.0 - 6.0). Participants were counted in the worst case category that their value changes to (low, normal or high), unless there is no change in their category. Participants whose laboratory value category was unchanged (e.g., High to High), or whose value became normal, were recorded in the "To Normal or No Change" category.
Time Frame: Up to 25 days
Population: Safety Population
Measure: Count of Participants; unit: Participants
Arm/Group | Part 2: Placebo | Part 2: GSK2838232 500 mg Tablet Fed
Number analyzed (Participants) | 3 | 7
Participants
  Glucose; To Low | 0 | 0
  Glucose; To Normal or No Change | 3 | 7
  Glucose; To High | 0 | 0
  Glucose; To Abnormal | 0 | 0
  Ketones; To Low | 0 | 0
  Ketones; To Normal or No Change | 3 | 7
  Ketones; To High | 0 | 0
  Ketones; To Abnormal | 0 | 0
  Occult blood; To Low | 0 | 0
  Occult blood; To Normal or No Change | 2 | 6
  Occult blood; To High | 0 | 0
  Occult blood; To Abnormal | 1 | 1
  Protein; To Low | 0 | 0
  Protein; To Normal or No Change | 3 | 7
  Protein; To High | 0 | 0
  Protein; To Abnormal | 0 | 0
  Specific gravity; To Low | 1 | 0
  Specific gravity; To Normal or No Change | 2 | 7
  Specific gravity; To High | 0 | 0
  Specific gravity; To Abnormal | 0 | 0
  Urine pH; To Low | 0 | 0
  Urine pH; To Normal or No Change | 3 | 7
  Urine pH; To High | 0 | 0
  Urine pH; To Abnormal | 0 | 0

10. Primary Outcome: Part 2: Blood Pressure at Indicated Time Points
Description: Systolic blood pressure (SBP) and diastolic blood pressure (DBP) were measured in supine position after 10 minutes rest for the participants at indicated time points.
Time Frame: Day -1; Pre-dose, 1, 4 hours on Day 1; 24 hours (Day 2); 48 hours (Day 3); 72 hours (Day 4), Days 5, 6, 7, 8, 9, 10; Pre-dose, 1, 4 , 24, 48, 72 hours on Day 11; Follow-up (Day 25)
Population: Safety Population
Measure: Mean (Standard Deviation); unit: Millimeter of mercury
Arm/Group | Part 2: Placebo | Part 2: GSK2838232 500 mg Tablet Fed
Number analyzed (Participants) | 3 | 7
Millimeter of mercury
  DBP; DAY -1 | 73.667 (7.5056) | 73.143 (4.7759)
  DBP; DAY 1, PREDOSE | 65.443 (2.6925) | 72.333 (8.1636)
  DBP; DAY 1, 1 Hour | 54.667 (3.7859) | 64.714 (5.8228)
  DBP; DAY 1, 4 Hours | 62.000 (1.0000) | 63.714 (6.7507)
  DBP; DAY 2, 24 Hours | 73.667 (4.0415) | 73.714 (6.0474)
  DBP; DAY 3, 48 Hours | 66.000 (1.7321) | 68.000 (7.3485)
  DBP; DAY 4, 72 Hours | 69.000 (2.6458) | 65.143 (8.3552)
  DBP; DAY 5 | 62.333 (4.9329) | 65.000 (7.3258)
  DBP; DAY 6 | 62.667 (4.5092) | 66.143 (6.6690)
  DBP; DAY 7 | 64.333 (3.0551) | 67.286 (4.8892)
  DBP; DAY 8 | 66.000 (2.6458) | 69.286 (6.3957)
  DBP; DAY 9 | 69.000 (4.0000) | 66.714 (5.0568)
  DBP; DAY 10 | 65.000 (7.2111) | 66.571 (8.0593)
  DBP; DAY 11, PREDOSE | 65.333 (5.1316) | 67.000 (8.0179)
  DBP; DAY 11, 1 Hour | 62.667 (7.3711) | 66.571 (7.6563)
  DBP; DAY 11, 4 Hours | 63.333 (4.5092) | 65.571 (8.5021)
  DBP; DAY 11, 24 Hours | 67.667 (4.5092) | 64.714 (7.0643)
  DBP; DAY 11, 48 Hours | 66.000 (5.5678) | 68.000 (8.9815)
  DBP; DAY 11, 72 Hours | 66.333 (3.7859) | 65.000 (5.8878)
  DBP; Follow-Up (DAY 25) | 71.000 (1.0000) | 76.143 (10.5424)
  SBP; DAY -1 | 121.000 (4.5826) | 123.000 (7.3258)
  SBP; DAY 1, PREDOSE | 107.553 (4.1400) | 121.190 (10.8374)
  SBP; DAY 1, 1 Hour | 99.333 (2.0817) | 113.000 (8.7178)
  SBP; DAY 1, 4 Hours | 105.000 (8.1854) | 106.286 (9.6214)
  SBP; DAY 2, 24 Hours | 110.667 (7.7675) | 113.286 (5.0568)
  SBP; DAY 3, 48 Hours | 111.333 (2.3094) | 111.714 (8.7695)
  SBP; DAY 4, 72 Hours | 108.333 (7.6376) | 109.000 (8.2260)
  SBP; DAY 5 | 105.667 (2.3094) | 109.000 (3.0551)
  SBP; DAY 6 | 106.667 (4.7258) | 107.857 (9.0079)
  SBP; DAY 7 | 103.333 (1.1547) | 112.143 (8.6106)
  SBP; DAY 8 | 105.667 (4.1633) | 109.571 (6.2412)
  SBP; DAY 9 | 107.333 (7.2342) | 110.143 (8.7069)
  SBP; DAY 10 | 110.000 (4.0000) | 106.714 (8.8828)
  SBP; DAY 11, PREDOSE | 107.113 (3.8626) | 110.333 (9.7088)
  SBP; DAY 11, 1 Hour | 113.000 (3.4641) | 111.571 (15.7041)
  SBP; DAY 11, 4 Hours | 108.667 (6.0277) | 109.857 (8.7069)
  SBP; DAY 11, 24 Hours | 107.333 (13.2035) | 105.143 (7.7337)
  SBP; DAY 11, 48 Hours | 109.667 (8.0829) | 109.286 (8.8828)
  SBP; DAY 11, 72 Hours | 110.333 (2.3094) | 110.286 (7.6966)
  SBP; Follow-Up (DAY 25) | 115.667 (5.8595) | 123.714 (10.6413)

11. Primary Outcome: Part 2: Change From Baseline in Blood Pressure
Description: SBP and DBP were measured in supine position after 10 minutes rest for participants at indicated time points. Baseline was defined as the latest pre-dose assessment, including those from unscheduled visits. Change from Baseline was defined as any visit value minus Baseline value.
Time Frame: Baseline (Day -1) and 1, 4 hours on Day 1; 24 hours (Day 2); 48 hours (Day 3); 72 hours (Day 4), Days 5, 6, 7, 8, 9, 10; Pre-dose, 1, 4 , 24, 48, 72 hours on Day 11; Follow-up (Day 25)
Population: Safety Population
Measure: Mean (Standard Deviation); unit: Millimeter of mercury
Arm/Group | Part 2: Placebo | Part 2: GSK2838232 500 mg Tablet Fed
Number analyzed (Participants) | 3 | 7
Millimeter of mercury
  DBP; DAY 1, 1 Hour | -10.777 (4.6690) | -7.619 (4.9086)
  DBP; DAY 1, 4 Hours | -3.443 (3.6851) | -8.619 (9.3099)
  DBP; DAY 2, 24 Hours | 8.223 (2.5455) | 1.381 (5.6866)
  DBP; DAY 3, 48 Hours | 0.557 (4.3485) | -4.333 (8.5244)
  DBP; DAY 4, 72 Hours | 3.557 (2.2180) | -7.190 (8.9524)
  DBP; DAY 5 | -3.110 (2.8366) | -7.333 (10.9039)
  DBP; DAY 6 | -2.777 (3.7175) | -6.190 (7.8255)
  DBP; DAY 7 | -1.110 (4.4381) | -5.047 (8.9388)
  DBP; DAY 8 | 0.557 (0.5095) | -3.047 (9.4939)
  DBP; DAY 9 | 3.557 (5.5901) | -5.619 (8.5770)
  DBP; DAY 10 | -0.443 (5.3488) | -5.761 (10.0756)
  DBP; DAY 11, PREDOSE | -0.110 (3.4708) | -5.333 (11.3081)
  DBP; DAY 11, 1 Hour | -2.777 (5.3385) | -5.761 (12.2366)
  DBP; DAY 11, 4 Hours | -2.110 (3.3729) | -6.761 (10.3364)
  DBP; DAY 11, 24 Hours | 2.223 (5.9279) | -7.619 (10.1445)
  DBP; DAY 11, 48 Hours | 0.557 (6.7022) | -4.333 (9.7243)
  DBP; DAY 11, 72 Hours | 0.890 (4.6224) | -7.333 (9.2678)
  DBP; Follow-Up (DAY 25) | 5.557 (3.2015) | 3.810 (10.1939)
  SBP; DAY 1, 1 Hour | -8.220 (3.0060) | -8.190 (10.8776)
  SBP; DAY 1, 4 Hours | -2.553 (5.6718) | -14.904 (8.2260)
  SBP; DAY 2, 24 Hours | 3.113 (5.8232) | -7.904 (8.7636)
  SBP; DAY 3, 48 Hours | 3.780 (1.8347) | -9.476 (6.2626)
  SBP; DAY 4, 72 Hours | 0.780 (5.4181) | -12.190 (7.1567)
  SBP; DAY 5 | -1.887 (3.6851) | -12.190 (11.9632)
  SBP; DAY 6 | -0.887 (7.0661) | -13.333 (15.5386)
  SBP; DAY 7 | -4.220 (3.7452) | -9.047 (13.8084)
  SBP; DAY 8 | -1.887 (5.1225) | -11.619 (11.8726)
  SBP; DAY 9 | -0.220 (6.1657) | -11.047 (14.9222)
  SBP; DAY 10 | 2.447 (7.8192) | -14.476 (13.8688)
  SBP; DAY 11, PREDOSE | -0.440 (4.4381) | -10.857 (13.9763)
  SBP; DAY 11, 1 Hour | 5.447 (6.6678) | -9.619 (19.6856)
  SBP; DAY 11, 4 Hours | 1.113 (2.6962) | -11.333 (14.3479)
  SBP; DAY 11, 24 Hours | -0.220 (13.2912) | -16.047 (15.2791)
  SBP; DAY 11, 48 Hours | 2.113 (12.0648) | -11.904 (11.8344)
  SBP; DAY 11, 72 Hours | 2.780 (1.8347) | -10.904 (13.1590)
  SBP; Follow-Up (DAY 25) | 8.113 (4.6808) | 2.524 (10.1553)

12. Primary Outcome: Part 2: Pulse Rate at Indicated Time Points
Description: Pulse rate of participants was measured in supine position after 10 minutes rest at indicated time points.
Time Frame: as for outcome 10
Population: Safety Population
Measure: Mean (Standard Deviation); unit: Beats per minute
Arm/Group | Part 2: Placebo | Part 2: GSK2838232 500 mg Tablet Fed
Number analyzed (Participants) | 3 | 7
Beats per minute
  DAY -1 | 63.667 (12.4231) | 64.143 (11.7817)
  DAY 1, PREDOSE | 63.663 (4.0415) | 63.714 (11.3991)
  DAY 1, 1 Hour | 68.000 (8.5440) | 72.286 (7.5214)
  DAY 1, 4 Hours | 64.667 (3.0551) | 66.000 (10.1160)
  DAY 2, 24 Hours | 57.667 (2.8868) | 58.286 (8.7123)
  DAY 3, 48 Hours | 58.000 (2.6458) | 59.429 (7.9762)
  DAY 4, 72 Hours | 58.667 (1.1547) | 58.286 (7.7613)
  DAY 5 | 60.667 (2.5166) | 66.429 (10.3900)
  DAY 6 | 62.333 (2.3094) | 59.143 (6.2564)
  DAY 7 | 59.333 (3.7859) | 63.429 (11.4143)
  DAY 8 | 64.333 (4.0415) | 62.000 (8.6795)
  DAY 9 | 61.000 (2.6458) | 60.714 (6.9693)
  DAY 10 | 63.667 (3.5119) | 60.143 (8.4346)
  DAY 11, PREDOSE | 61.887 (1.3891) | 60.810 (9.3355)
  DAY 11, 1 Hour | 72.667 (4.7258) | 70.143 (7.0102)
  DAY 11, 4 Hours | 68.000 (5.2915) | 68.857 (8.4148)
  DAY 11, 24 Hours | 67.667 (6.4291) | 64.571 (7.3679)
  DAY 11, 48 Hours | 61.667 (6.5064) | 61.714 (4.6085)
  DAY 11, 72 Hours | 63.000 (2.6458) | 60.857 (3.9340)
  Follow-Up (DAY 25) | 70.667 (8.0829) | 63.857 (9.4062)

13. Primary Outcome: Part 2: Change From Baseline in Pulse Rate
Description: Pulse rate was measured in supine position after 10 minutes rest at indicated time points. Baseline was defined as the latest pre-dose assessment, including those from unscheduled visits. Change from Baseline was defined as any visit value minus Baseline value.
Time Frame: as for outcome 11
Population: Safety Population
Measure: Mean (Standard Deviation); unit: Beats per minute
Arm/Group | Part 2: Placebo | Part 2: GSK2838232 500 mg Tablet Fed
Number analyzed (Participants) | 3 | 7
Beats per minute
  DAY 1, 1 Hour | 4.337 (11.2398) | 8.571 (5.4337)
  DAY 1, 4 Hours | 1.003 (6.6583) | 2.286 (9.4965)
  DAY 2, 24 Hours | -5.997 (2.5166) | -5.429 (4.4808)
  DAY 3, 48 Hours | -5.663 (4.9329) | -4.286 (5.9568)
  DAY 4, 72 Hours | -4.997 (5.1316) | -5.429 (7.0937)
  DAY 5 | -2.997 (5.6862) | 2.714 (11.2383)
  DAY 6 | -1.330 (4.3589) | -4.571 (9.8771)
  DAY 7 | -4.330 (1.0000) | -0.286 (12.4265)
  DAY 8 | 0.670 (0.0000) | -1.714 (8.2357)
  DAY 9 | -2.663 (4.9329) | -3.000 (9.7265)
  DAY 10 | 0.003 (7.5056) | -3.571 (10.5886)
  DAY 11, PREDOSE | -1.777 (4.1400) | -2.904 (10.5699)
  DAY 11, 1 Hour | 9.003 (8.3865) | 6.429 (10.3760)
  DAY 11, 4 Hours | 4.337 (8.5049) | 5.143 (10.9028)
  DAY 11, 24 Hours | 4.003 (6.5064) | 0.857 (10.2185)
  DAY 11, 48 Hours | -1.997 (9.4516) | -2.000 (9.6686)
  DAY 11, 72 Hours | -0.663 (4.0415) | -2.857 (8.7974)
  Follow-Up (DAY 25) | 7.003 (11.9304) | 0.143 (10.7995)

14. Primary Outcome: Part 2: Number of Participants With Abnormal Electrocardiogram (ECG) Findings
Description: Single and triplicate 12-lead ECG's were obtained at least 5 minutes apart in the supine position after 10 minutes of rest at indicated time points using an ECG machine that automatically calculates the heart rate and measures PR, QRS, QT and QT duration corrected for heart rate by Fridericia's formula (QTcF) intervals. Clinically significant (CS) and not clinically significant (NCS) abnormal ECG findings have been presented. CS abnormal findings are those which are not associated with the underlying disease, unless judged by the investigator to be more severe than expected for the participant's condition.
Time Frame: Day -1; 1, 4, 12 hours on Day 1; Days 2, 3, 5, 8; 1, 4, 12, 24 Hours on Day 11; Follow-up (Day 25)
Population: Safety Population
Measure: Count of Participants; unit: Participants
Arm/Group | Part 2: Placebo | Part 2: GSK2838232 500 mg Tablet Fed
Number analyzed (Participants) | 3 | 7
Participants
  NCS: DAY -1 | 2 | 6
  CS: DAY -1 | 0 | 0
  NCS: DAY 1, 1 Hour | 2 | 4
  CS: DAY 1, 1 Hour | 0 | 0
  NCS: DAY 1, 4 Hours | 2 | 6
  CS: DAY 1, 4 Hours | 0 | 0
  NCS: DAY 1, 12 Hours | 3 | 6
  CS: DAY 1, 12 Hours | 0 | 0
  NCS: DAY 2 | 2 | 5
  CS: DAY 2 | 0 | 0
  NCS: DAY 3 | 3 | 5
  CS: DAY 3 | 0 | 0
  NCS: DAY 5 | 3 | 6
  CS: DAY 5 | 0 | 0
  NCS: DAY 8 | 2 | 7
  CS: DAY 8 | 0 | 0
  NCS: DAY 11, 1 Hour | 2 | 3
  CS: DAY 11, 1 Hour | 0 | 0
  NCS: DAY 11, 4 Hours | 2 | 5
  CS: DAY 11, 4 Hours | 0 | 0
  NCS: DAY 11, 12 Hours | 2 | 4
  CS: DAY 11, 12 Hours | 0 | 0
  NCS: DAY 11, 24 Hours | 2 | 5
  CS: DAY 11, 24 Hours | 0 | 0
  NCS: Follow-up (DAY 25) | 1 | 6
  CS: Follow-up (DAY 25) | 0 | 0

15. Primary Outcome: Part 2: Change From Baseline in Mean Heart Rate Values as ECG Parameter
Description: Single and triplicate 12-lead ECG's were obtained at least 5 minutes apart in the supine position after 10 minutes of rest at indicated time points using an ECG machine that automatically calculates the heart rate. Baseline was defined as the latest pre-dose assessment, including those from unscheduled visits. Change from Baseline was defined as any visit value minus Baseline value.
Time Frame: Baseline (Day -1) and 1, 4, 12 hours on Day 1; Days 2, 3 5, 8; Pre-dose, 1, 4, 12, 24 hours Day 11; Follow-up (Day 25)
Population: Safety Population
Measure: Mean (Standard Deviation); unit: Beats per minute
Arm/Group | Part 2: Placebo | Part 2: GSK2838232 500 mg Tablet Fed
Number analyzed (Participants) | 3 | 7
Beats per minute
  DAY 1, 1 Hour | 4.000 (10.1734) | 10.240 (5.0930)
  DAY 1, 4 Hours | 2.000 (5.9287) | 1.954 (3.9733)
  DAY 1, 12 Hours | -6.000 (6.8912) | 0.526 (5.1336)
  DAY 2 | -8.000 (0.8826) | -5.331 (4.8861)
  DAY 3 | -5.333 (5.4902) | -1.046 (4.9332)
  DAY 5 | -3.667 (2.6062) | 2.669 (11.9804)
  DAY 8 | -2.000 (1.8571) | 0.954 (5.8978)
  DAY 11, PREDOSE | -4.333 (1.7670) | -0.903 (6.9388)
  DAY 11, 1 Hour | 10.333 (7.7564) | 6.383 (5.9634)
  DAY 11, 4 Hours | 1.000 (4.0986) | 4.811 (8.2683)
  DAY 11, 12 Hours | -0.667 (3.8461) | -0.189 (5.6490)
  DAY 11, 24 Hours | 2.667 (4.8106) | 0.954 (4.8878)
  Follow-up (DAY 25) | 2.333 (12.4705) | 0.669 (8.2733)

16. Primary Outcome: Part 2: Change From Baseline in PR Interval, QRS, QT Interval, and QTcF Interval as ECG Parameters
Description: Single and triplicate 12-lead ECG's were obtained at least 5 minutes apart in the supine position after 10 minutes of rest at indicated time points using an ECG machine that automatically calculates measures PR, QRS, QT and QTcF intervals. Baseline was defined as the latest pre-dose assessment, including those from unscheduled visits. Change from Baseline was defined as any visit value minus Baseline value.
Time Frame: Baseline (Day -1) and 1, 4, 12 hours on Day 1; Days 2, 3 5, 8; Pre-dose, 1, 4, 12, 24 hours Day 11; Follow-up (Day 25)
Population: Safety Population
Measure: Mean (Standard Deviation); unit: Milliseconds
Arm/Group | Part 2: Placebo | Part 2: GSK2838232 500 mg Tablet Fed
Number analyzed (Participants) | 3 | 7
Milliseconds
  PR interval; DAY 1, 1 Hour | -7.110 (2.0360) | -3.999 (10.6110)
  PR interval; DAY 1, 4 Hours | -6.443 (3.7945) | -12.284 (13.9800)
  PR interval; DAY 1, 12 Hours | -0.443 (11.9348) | 3.430 (5.7511)
  PR interval; DAY 2 | 4.890 (3.6695) | 3.716 (5.1471)
  PR interval; DAY 3 | 1.557 (4.2847) | 4.573 (6.1252)
  PR interval; DAY 5 | 6.223 (9.1999) | 2.287 (9.5818)
  PR interval; DAY 8 | 6.223 (10.8609) | 7.430 (11.6897)
  PR interval; DAY 11, PREDOSE | 5.113 (10.1172) | 7.620 (5.5483)
  PR interval; DAY 11, 1 Hour | -5.777 (7.3456) | 2.287 (5.2749)
  PR interval; DAY 11, 4 Hours | -3.110 (10.8418) | -0.570 (9.9657)
  PR interval; DAY 11, 12 Hours | 4.223 (12.6221) | 1.716 (9.4661)
  PR interval; DAY 11, 24 Hours | 2.890 (10.8418) | 3.144 (6.0321)
  PR interval; Follow-up (DAY 25) | -10.443 (5.0039) | 2.001 (13.1373)
  QRS interval; DAY 1, 1 Hour | 3.330 (5.2915) | -1.713 (3.3072)
  QRS interval; DAY 1, 4 Hours | 1.997 (4.6188) | -1.713 (1.4322)
  QRS interval; DAY 1, 12 Hours | 6.663 (4.6188) | 1.716 (3.6295)
  QRS interval; DAY 2 | 1.330 (2.0000) | 0.287 (2.2711)
  QRS interval; DAY 3 | 2.663 (3.0551) | -4.570 (5.8288)
  QRS interval; DAY 5 | 3.997 (4.1633) | -1.999 (2.8532)
  QRS interval; DAY 8 | -0.003 (1.1547) | -3.141 (4.1578)
  QRS interval; DAY 11, PREDOSE | 1.107 (4.3393) | -0.570 (1.9401)
  QRS interval; DAY 11, 1 Hour | -0.003 (2.3094) | -0.856 (5.1594)
  QRS interval; DAY 11, 4 Hours | -1.337 (1.1547) | -2.570 (3.0890)
  QRS interval; DAY 11, 12 Hours | 3.330 (3.4641) | -0.856 (4.4676)
  QRS interval; DAY 11, 24 Hours | -1.337 (1.1547) | -0.570 (3.7401)
  QRS interval; Follow-up (DAY 25) | 1.997 (11.0151) | 1.716 (1.5811)
  QT interval; DAY 1, 1 Hour | -8.223 (18.0177) | -26.094 (12.8322)
  QT interval; DAY 1, 4 Hours | -3.557 (9.7159) | -11.523 (11.6047)
  QT interval; DAY 1, 12 Hours | 18.443 (18.0654) | -7.237 (15.5856)
  QT interval; DAY 2 | 5.777 (4.0741) | 0.763 (9.3458)
  QT interval; DAY 3 | 5.777 (18.7403) | -8.951 (11.9189)
  QT interval; DAY 5 | -0.890 (8.9502) | -10.666 (19.1883)
  QT interval; DAY 8 | 1.110 (2.3378) | -8.951 (14.2945)
  QT interval; DAY 11, PREDOSE | 5.553 (6.1963) | -4.283 (13.7560)
  QT interval; DAY 11, 1 Hour | -18.223 (12.2979) | -28.380 (19.3087)
  QT interval; DAY 11, 4 Hours | -8.223 (10.0299) | -20.380 (17.7740)
  QT interval; DAY 11, 12 Hours | 5.777 (10.5451) | -13.237 (13.1751)
  QT interval; DAY 11, 24 Hours | -10.890 (12.6010) | -13.523 (11.7381)
  QT interval; Follow-up (DAY 25) | 0.443 (26.9777) | -3.237 (20.6284)
  QTcF interval; DAY 1, 1 Hour | -0.667 (6.3366) | -5.857 (10.3146)
  QTcF interval; DAY 1, 4 Hours | 1.000 (2.1838) | -7.429 (7.1165)
  QTcF interval; DAY 1, 12 Hours | 7.000 (8.2158) | -6.286 (10.9182)
  QTcF interval; DAY 2 | -10.667 (4.6671) | -10.143 (6.7366)
  QTcF interval; DAY 3 | -5.000 (7.6908) | -10.714 (9.6264)
  QTcF interval; DAY 5 | -7.667 (4.1800) | -6.286 (7.6605)
  QTcF interval; DAY 8 | -2.000 (2.0246) | -6.714 (6.5305)
  QTcF interval; DAY 11, PREDOSE | -2.887 (2.9150) | -6.476 (5.7033)
  QTcF interval; DAY 11, 1 Hour | 1.000 (4.8434) | -15.286 (11.1814)
  QTcF interval; DAY 11, 4 Hours | -5.667 (6.1719) | -11.000 (4.8767)
  QTcF interval; DAY 11, 12 Hours | 5.333 (3.8474) | -12.571 (7.6845)
  QTcF interval; DAY 11, 24 Hours | -5.667 (2.9652) | -10.429 (7.7286)
  QTcF interval; Follow-up (DAY 25) | 4.000 (5.8145) | -2.571 (12.9581)

17. Primary Outcome: Part 2: Area Under the Plasma Drug Concentration Time Curve From Pre-dose to the End of the Dosing Interval at Steady State (AUC[0-tau]) Following Administration of Non-boosted Once-daily Doses of GSK2838232 Tablet in Fed State
Description: Blood samples were collected at indicated time points for pharmacokinetic analysis of GSK2838232 given as a non-boosted once-daily dosing tablet in fed state. Pharmacokinetic parameters were determined using standard non-compartmental methods.
Time Frame: Pre-dose, 0.5,1, 1.5, 2, 2.5, 3, 3.5, 4, 6, 8, 12 and 24 hours post-dose on Day 1; Pre-dose, 0.5, 1, 1.5, 2, 2.5, 3, 3.5, 4, 6, 8, 12, 24, 36, 48, 72, 96 and 120 hours post-dose on Day 11 in Part 2
Population: Pharmacokinetic Population
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: Hours*nanograms per milliliter
Arm/Group | Part 2: GSK2838232 500 mg Tablet Fed
Number analyzed (Participants) | 7
Hours*nanograms per milliliter
  Day 1 | 895.42 (39.08)
  Day 11 | 1184.55 (35.34)

18. Primary Outcome: Part 2: Cmax Following Administration of Non-boosted Once-daily Doses of GSK2838232 Tablet in Fed State
Description: as for outcome 17
Time Frame: as for outcome 17
Population: Pharmacokinetic Population
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: Nanograms per milliliter
Arm/Group | Part 2: GSK2838232 500 mg Tablet Fed
Number analyzed (Participants) | 7
Nanograms per milliliter
  Day 1 | 79.575 (45.69)
  Day 11 | 94.239 (34.24)

19. Primary Outcome: Part 2: Observed Concentration at the End of the Dosing Interval (Ctau) Following Administration of Non-boosted Once-daily Doses of GSK2838232 Tablet in Fed State
Description: as for outcome 17
Time Frame: as for outcome 17
Population: Pharmacokinetic Population
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: Nanograms per milliliter
Arm/Group | Part 2: GSK2838232 500 mg Tablet Fed
Number analyzed (Participants) | 7
Nanograms per milliliter
  Day 1 | 21.620 (42.51)
  Day 11 | 27.668 (41.16)

20. Primary Outcome: Part 2: Tmax Following Administration of Non-boosted Once-daily Doses of GSK2838232 Tablet in Fed State
Description: as for outcome 17
Time Frame: as for outcome 17
Population: Pharmacokinetic Population
Measure: Median (Full Range); unit: Hours
Arm/Group | Part 2: GSK2838232 500 mg Tablet Fed
Number analyzed (Participants) | 7
Hours
  Day 1 | 4.000 [2.00 to 8.00]
  Day 11 | 3.500 [1.98 to 6.00]

21. Primary Outcome: Part 2: Lag-time (Tlag) Following Administration of Non-boosted Once-daily Doses of GSK2838232 Tablet in Fed State on Day 1
Description: Blood samples were collected at indicated time points for pharmacokinetic analysis of GSK2838232 given as a non-boosted once-daily dosing tablet in fed state. Tlag is a time delay between drug administration and first observed concentration. Pharmacokinetic parameters were determined using standard non-compartmental methods.
Time Frame: Pre-dose, 0.5,1, 1.5, 2, 2.5, 3, 3.5, 4, 6, 8, 12 and 24 hours post-dose on Day 1 in Part 2
Population: Pharmacokinetic Population
Measure: Median (Full Range); unit: Hours
Arm/Group | Part 2: GSK2838232 500 mg Tablet Fed
Number analyzed (Participants) | 7
Hours | 0.500 [0.00 to 1.00]

22. Primary Outcome: Part 2: AUC(0-infinity) Following Administration of Non-boosted Once-daily Doses of GSK2838232 Tablet in Fed State on Day 11
Description: as for outcome 17
Time Frame: Pre-dose, 0.5, 1, 1.5, 2, 2.5, 3, 3.5, 4, 6, 8, 12, 24, 36, 48, 72, 96 and 120 hours post-dose on Day 11 in Part 2
Population: Pharmacokinetic Population
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: Hours*nanograms per milliliter
Arm/Group | Part 2: GSK2838232 500 mg Tablet Fed
Number analyzed (Participants) | 7
Hours*nanograms per milliliter | 1816.34 (37.32)

23. Primary Outcome: Part 2: Apparent Terminal Phase Half-life (T1/2) Following Administration of Non-boosted Once-daily Doses of GSK2838232 Tablet in Fed State on Day 11
Description: as for outcome 17
Time Frame: Pre-dose, 0.5, 1, 1.5, 2, 2.5, 3, 3.5, 4, 6, 8, 12, 24, 36, 48, 72, 96 and 120 hours post-dose on Day 11 in Part 2
Population: Pharmacokinetic Population
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: Hours
Arm/Group | Part 2: GSK2838232 500 mg Tablet Fed
Number analyzed (Participants) | 7
Hours | 23.217 (37.85)

24. Primary Outcome: Part 2: Time of Last Quantifiable Concentration (Tlast) Following Administration of Non-boosted Once-daily Doses of GSK2838232 Tablet in Fed State on Day 11
Description: as for outcome 17
Time Frame: Pre-dose, 0.5, 1, 1.5, 2, 2.5, 3, 3.5, 4, 6, 8, 12, 24, 36, 48, 72, 96 and 120 hours post-dose on Day 11 in Part 2
Population: Pharmacokinetic Population
Measure: Median (Full Range); unit: Hours
Arm/Group | Part 2: GSK2838232 500 mg Tablet Fed
Number analyzed (Participants) | 7
Hours | 118.800 [95.10 to 118.85]

25. Secondary Outcome: Part 1: Number of Participants With SAEs and Non-SAEs
Description: An AE is any untoward medical occurrence in a clinical study participant, temporally associated with the use of a study treatment, whether or not considered related to the study treatment. SAE is defined as any untoward medical occurrence that, at any dose results in death, is life threatening, requires hospitalization or prolongation of existing hospitalization, results in persistent disability/incapacity, is a congenital anomaly/ birth defect, is associated with liver injury or impaired liver function or any other situations as per medical or scientific judgment. Number of participants with SAEs and common non-SAEs (>=5%) are presented.
Time Frame: Up to 60 days
Population: Safety Population
Measure: Count of Participants; unit: Participants
Arm/Group | Part 1: GSK2838232 200 mg/Ritonavir Capsule Fed | Part 1: GSK2838232 200 mg/Ritonavir Tablet Fed | Part 1: GSK2838232 200 mg/Ritonavir Tablet Fasted
Number analyzed (Participants) | 15 | 15 | 14
Participants
  Any SAE | 0 | 0 | 0
  Any non-SAE | 3 | 2 | 1

26. Secondary Outcome: Part 1: Number of Participants With Worst Case Hematology Results to PCI Criteria
Description: Blood samples were collected from participants for analysis of following hematology parameters; hematocrit, hemoglobin, leukocytes, lymphocytes, neutrophils and platelets. PCI ranges were >0.54 as proportion of red blood cells in blood for hematocrit, >180 g/L for hemoglobin, < 3 or >20 cells/L for leukocytes, 0.8 x10^9 cells/L for lymphocytes, 1.5 x10^9 cells/L for neutrophils, and <100 or >550 cells/L for platelets. Participants were counted in the worst case category that their value changes to (low, within range or no change, or high), unless there is no change in their category. Participants whose laboratory value category was unchanged (e.g., High to High), or whose value became within range, were recorded in the "To within Range or No Change" category.
Time Frame: Up to 60 days
Population: Safety Population
Measure: Count of Participants; unit: Participants
Arm/Group | Part 1: GSK2838232 200 mg/Ritonavir Capsule Fed | Part 1: GSK2838232 200 mg/Ritonavir Tablet Fed | Part 1: GSK2838232 200 mg/Ritonavir Tablet Fasted
Number analyzed (Participants) | 15 | 15 | 14
Participants
  Hematocrit; To Low | 0 | 0 | 0
  Hematocrit; To within Range or No Change | 15 | 15 | 14
  Hematocrit; To High | 0 | 0 | 0
  Hemoglobin; To Low | 0 | 0 | 0
  Hemoglobin; To within Range or No Change | 15 | 15 | 14
  Hemoglobin; To High | 0 | 0 | 0
  Leukocytes; To Low | 0 | 0 | 0
  Leukocytes; To within Range or No Change | 15 | 15 | 14
  Leukocytes; To High | 0 | 0 | 0
  Lymphocytes; To Low | 0 | 0 | 0
  Lymphocytes; To within Range or No Change | 15 | 15 | 14
  Lymphocytes; To High | 0 | 0 | 0
  Neutrophils; To Low | 0 | 0 | 0
  Neutrophils; To within Range or No Change | 15 | 15 | 14
  Neutrophils; To High | 0 | 0 | 0
  Platelets; To Low | 0 | 0 | 0
  Platelets; To within Range or No Change | 15 | 15 | 14
  Platelets; To High | 0 | 0 | 0

27. Secondary Outcome: Part 1: Number of Participants With Worst Case Clinical Chemistry Results to PCI Criteria
Description: Blood samples were collected from participants for analysis of following clinical chemistry parameters; glucose, ALT, albumin, alkaline phosphatase, AST, bilirubin, calcium, potassium and sodium. PCI ranges were <30 g/L for albumin, <2 or 2.75 mmol/L for calcium, <3 or >9 mmol/L for glucose, >=2 times ULN U/L for ALT, >=2 times ULN U/L for alkaline phosphatase, >=2 times ULN U/L for AST, >=1.5 times ULN µmol/L for bilirubin, <3 or >5.5 mmol/L for potassium, and <130 or >150 mmol/L for sodium. Participants were counted in the worst case category that their value changes to (low, within range or no change,or high), unless there is no change in their category. Participants whose laboratory value category was unchanged (e.g., High to High), or whose value became within range, were recorded in the "To within Range or No Change" category.
Time Frame: Up to 60 days
Population: Safety Population
Measure: Count of Participants; unit: Participants
Arm/Group | Part 1: GSK2838232 200 mg/Ritonavir Capsule Fed | Part 1: GSK2838232 200 mg/Ritonavir Tablet Fed | Part 1: GSK2838232 200 mg/Ritonavir Tablet Fasted
Number analyzed (Participants) | 15 | 15 | 14
Participants
  Glucose; To Low | 0 | 0 | 0
  Glucose; To within Range or No Change | 15 | 15 | 14
  Glucose; To High | 0 | 0 | 0
  ALT; To Low | 0 | 0 | 0
  ALT; To within Range or No Change | 15 | 15 | 14
  ALT; To High | 0 | 0 | 0
  Albumin; To Low | 0 | 0 | 0
  Albumin; To within Range or No Change | 15 | 15 | 14
  Albumin; To High | 0 | 0 | 0
  Alkaline phosphatase; To Low | 0 | 0 | 0
  Alkaline phosphatase; To within Range or No Change | 15 | 15 | 14
  Alkaline phosphatase; To High | 0 | 0 | 0
  AST; To Low | 0 | 0 | 0
  AST; To within Range or No Change | 15 | 15 | 14
  AST; To High | 0 | 0 | 0
  Bilirubin; To Low | 0 | 0 | 0
  Bilirubin; To within Range or No Change | 15 | 15 | 14
  Bilirubin; To High | 0 | 0 | 0
  Calcium; To Low | 0 | 0 | 0
  Calcium; To within Range or No Change | 15 | 15 | 14
  Calcium; To High | 0 | 0 | 0
  Potassium; To Low | 0 | 0 | 0
  Potassium; To within Range or No Change | 15 | 15 | 14
  Potassium; To High | 0 | 0 | 0
  Sodium; To Low | 0 | 0 | 0
  Sodium; To within Range or No Change | 15 | 15 | 14
  Sodium; To High | 0 | 0 | 0

28. Secondary Outcome: Part 1: Number of Participants With Worst Case Urinalysis Results Relative to Normal Range Criteria
Description: Urine samples were collected from participants for analysis of following urinalysis parameters; specific gravity, pH, presence of glucose, protein, occult blood, ketones in urine analyzed by dipstick method. The dipstick test gives results in a semi-quantitative manner. Urine specific gravity is a measure of the concentration of solutes in the urine and provides information on the kidney's ability to concentrate urine. The reference range is 1.002-1.030. Urine pH is an acid-base measurement. Normal urine has a slightly acid pH (5.0 - 6.0). Participants were counted in the worst case category that their value changes to (low, normal or high), unless there is no change in their category. Participants whose laboratory value category was unchanged (e.g., High to High), or whose value became normal, were recorded in the "To Normal or No Change" category.
Time Frame: Up to 60 days
Population: Safety Population
Measure: Count of Participants; unit: Participants
Arm/Group | Part 1: GSK2838232 200 mg/Ritonavir Capsule Fed | Part 1: GSK2838232 200 mg/Ritonavir Tablet Fed | Part 1: GSK2838232 200 mg/Ritonavir Tablet Fasted
Number analyzed (Participants) | 15 | 15 | 14
Participants
  Glucose; To Low | 0 | 0 | 0
  Glucose; To Normal or No Change | 15 | 15 | 14
  Glucose; To High | 0 | 0 | 0
  Glucose; To Abnormal | 0 | 0 | 0
  Ketones; To Low | 0 | 0 | 0
  Ketones; To Normal or No Change | 14 | 15 | 14
  Ketones; To High | 0 | 0 | 0
  Ketones To Abnormal | 1 | 0 | 0
  Occult blood; To Low | 0 | 0 | 0
  Occult blood ; To Normal or No Change | 14 | 13 | 10
  Occult blood; To High | 0 | 0 | 0
  Occult blood To Abnormal | 1 | 2 | 4
  Protein; To Low | 0 | 0 | 0
  Protein; To Normal or No Change | 15 | 15 | 14
  Protein; To High | 0 | 0 | 0
  Protein To Abnormal | 0 | 0 | 0
  Specific gravity; To Low | 1 | 0 | 2
  Specific gravity; To Normal or No Change | 14 | 15 | 12
  Specific gravity; To High | 0 | 0 | 0
  Specific gravity To Abnormal | 0 | 0 | 0
  Urine pH; To Low | 0 | 0 | 0
  Urine pH; To Normal or No Change | 15 | 15 | 14
  Urine pH; To High | 0 | 0 | 0
  Urine pH; To Abnormal | 0 | 0 | 0

29. Secondary Outcome: Part 1: Blood Pressure at Indicated Time Points
Description: SBP and DBP of participants were measured in supine position after 10 minutes rest at indicated time points.
Time Frame: Day -2; Day -1; Pre-dose, 1, 2, 4, 6, 8, 12, 24, 48, 72 Hours on Day 1
Population: Safety Population
Measure: Mean (Standard Deviation); unit: Millimeter of mercury
Arm/Group | Part 1: GSK2838232 200 mg/Ritonavir Capsule Fed | Part 1: GSK2838232 200 mg/Ritonavir Tablet Fed | Part 1: GSK2838232 200 mg/Ritonavir Tablet Fasted
Number analyzed (Participants) | 15 | 15 | 14
Millimeter of mercury
  DBP; DAY -2 | 68.667 (6.2981) | 69.533 (7.6426) | 65.000 (6.1893)
  DBP; DAY -1 | 67.467 (6.2320) | 68.467 (8.7657) | 65.643 (7.7619)
  DBP; DAY 1, PREDOSE | 65.956 (4.9419) | 66.245 (7.1653) | 66.929 (7.4379)
  DBP; DAY 1, 1 Hour | 63.200 (6.1551) | 64.133 (6.1163) | 67.357 (5.4998)
  DBP; DAY 1, 2 Hours | 62.133 (5.6552) | 62.533 (4.6425) | 66.071 (7.1410)
  DBP; DAY 1, 4 Hours | 63.733 (6.6490) | 64.400 (5.3825) | 67.429 (5.5152)
  DBP; DAY 1, 6 Hours | 64.400 (6.1968) | 64.067 (7.4878) | 66.071 (5.5117)
  DBP; DAY 1, 8 Hours | 68.333 (6.6940) | 66.933 (5.0351) | 68.000 (6.1269)
  DBP; DAY 1, 12 Hours | 68.867 (5.5532) | 67.800 (7.2723) | 66.214 (5.1766)
  DBP; DAY 1, 24 Hours | 68.400 (6.4343) | 66.533 (6.2663) | 66.929 (7.0870)
  DBP; DAY 1, 48 Hours | 66.600 (7.4431) | 67.333 (5.5377) | 64.643 (6.1595)
  DBP; DAY 1, 72 Hours | 66.600 (8.0250) | 67.067 (5.2026) | 64.429 (7.1545)
  SBP; DAY -2 | 108.667 (9.9115) | 109.733 (9.0116) | 105.786 (9.8775)
  SBP; DAY -1 | 110.067 (10.2153) | 104.000 (9.7980) | 108.429 (11.1128)
  SBP; DAY 1, PREDOSE | 108.156 (9.2400) | 108.289 (11.1021) | 106.858 (9.5900)
  SBP; DAY 1, 1 Hour | 106.000 (10.0428) | 108.400 (8.3820) | 106.500 (9.3377)
  SBP; DAY 1, 2 Hours | 104.867 (10.6091) | 105.067 (9.6323) | 106.214 (11.8593)
  SBP; DAY 1, 4 Hours | 107.733 (9.1844) | 106.000 (8.8237) | 106.714 (10.8019)
  SBP; DAY 1, 6 Hours | 108.333 (8.9894) | 106.933 (7.1661) | 108.214 (11.8008)
  SBP; DAY 1, 8 Hours | 112.067 (8.9639) | 110.600 (12.3508) | 106.000 (12.3973)
  SBP; DAY 1, 12 Hours | 110.133 (10.2181) | 113.000 (11.9762) | 107.786 (12.1919)
  SBP; DAY 1, 24 Hours | 106.200 (9.9441) | 107.467 (10.8619) | 105.500 (11.1061)
  SBP; DAY 1, 48 Hours | 106.867 (10.1620) | 107.067 (6.3860) | 102.000 (12.2725)
  SBP; DAY 1, 72 Hours | 104.067 (11.7075) | 105.933 (10.8197) | 107.429 (13.5290)

30. Secondary Outcome: Part 1: Change From Baseline in Blood Pressure
Description: SBP and DBP were measured in supine position after 10 minutes rest for the participant at indicated time points. Baseline was defined as the latest pre-dose assessment, including those from unscheduled visits. Change from Baseline was defined as any visit value minus Baseline value.
Time Frame: Baseline (Day -1) and 1, 2, 4, 6, 8, 12, 24, 48, 72 Hours on Day 1
Population: Safety Population
Measure: Mean (Standard Deviation); unit: Millimeter of mercury
Arm/Group | Part 1: GSK2838232 200 mg/Ritonavir Capsule Fed | Part 1: GSK2838232 200 mg/Ritonavir Tablet Fed | Part 1: GSK2838232 200 mg/Ritonavir Tablet Fasted
Number analyzed (Participants) | 15 | 15 | 14
Millimeter of mercury
  DBP; DAY 1, 1 Hour | -2.756 (4.5583) | -2.112 (5.8242) | 0.429 (6.2950)
  DBP; DAY 1, 2 Hours | -3.823 (4.8274) | -3.712 (7.5868) | -0.857 (6.0936)
  DBP; DAY 1, 4 Hours | -2.223 (5.1037) | -1.845 (6.6186) | 0.500 (4.4191)
  DBP; DAY 1, 6 Hours | -1.556 (4.0795) | -2.179 (5.8416) | -0.857 (6.7412)
  DBP; DAY 1, 8 Hours | 2.377 (3.8999) | 0.688 (7.8368) | 1.071 (4.3963)
  DBP; DAY 1, 12 Hours | 2.911 (6.7287) | 1.555 (7.1028) | -0.714 (6.2782)
  DBP; DAY 1, 24 Hours | 2.444 (4.7072) | 0.288 (6.5408) | 0.000 (6.3519)
  DBP; DAY 1, 48 Hours | 0.644 (7.9350) | 1.088 (8.1406) | -2.286 (4.2171)
  DBP; DAY 1, 72 Hours | 0.644 (6.4814) | 0.821 (6.3773) | -2.500 (7.5579)
  SBP; DAY 1, 1 Hour | -2.156 (5.2225) | 0.111 (8.8653) | -0.358 (7.2826)
  SBP; DAY 1, 2 Hours | -3.289 (8.9001) | -3.222 (11.2680) | -0.644 (6.9132)
  SBP; DAY 1, 4 Hours | -0.423 (7.3588) | -2.289 (10.0523) | -0.144 (8.8536)
  SBP; DAY 1, 6 Hours | 0.177 (6.2989) | -1.355 (8.9097) | 1.356 (9.9739)
  SBP; DAY 1, 8 Hours | 3.911 (7.8095) | 2.311 (11.0679) | -0.858 (10.0987)
  SBP; DAY 1, 12 Hours | 1.977 (6.7186) | 4.711 (7.4998) | 0.928 (9.8279)
  SBP; DAY 1, 24 Hours | -1.956 (7.9095) | -0.822 (9.2810) | -1.358 (4.6289)
  SBP; DAY 1, 48 Hours | -1.289 (4.9058) | -1.222 (10.7458) | -4.858 (9.5294)
  SBP; DAY 1, 72 Hours | -4.089 (7.4727) | -2.355 (9.9198) | 0.571 (11.2671)

31. Secondary Outcome: Part 1: Pulse Rate at Indicated Time Points
Description: Pulse rate was measured in supine position after 10 minutes rest for the participant at indicated time points.
Time Frame: Day -2; Day -1; Pre-dose, 1, 2, 4, 6, 8, 12, 24, 48, 72 Hours on Day 1
Population: Safety Population
Measure: Mean (Standard Deviation); unit: Beats per minute
Groups:
- Part 1: GSK 200 mg/Ritonavir Tablet Fasted: Participants received a single dose of GSK2838232 200 mg (as 2 x 100 mg) tablet formulation under fasted conditions in treatment period 3 along with ritonavir 100 mg tablet to be taken with water in fasted condition.
Arm/Group | Part 1: GSK2838232 200 mg/Ritonavir Capsule Fed | Part 1: GSK2838232 200 mg/Ritonavir Tablet Fed | Part 1: GSK 200 mg/Ritonavir Tablet Fasted
Number analyzed (Participants) | 15 | 15 | 14
Beats per minute
  DAY -2 | 64.067 (14.6066) | 62.333 (10.8737) | 60.214 (9.4558)
  DAY -1 | 62.333 (10.6212) | 63.067 (7.6108) | 59.071 (10.6516)
  DAY 1, PREDOSE | 65.023 (10.7156) | 64.311 (7.9777) | 59.857 (8.3402)
  DAY 1, 1 Hour | 74.667 (8.5996) | 72.333 (9.2711) | 58.571 (9.3949)
  DAY 1, 2 Hours | 72.667 (11.8301) | 72.933 (9.5877) | 60.214 (10.4010)
  DAY 1, 4 Hours | 68.133 (7.8728) | 69.467 (11.0574) | 61.214 (9.5287)
  DAY 1, 6 Hours | 68.867 (9.9417) | 68.133 (11.0961) | 66.500 (9.4360)
  DAY 1, 8 Hours | 66.533 (10.5144) | 66.933 (7.2552) | 63.571 (10.6027)
  DAY 1, 12 Hours | 64.867 (9.0069) | 65.867 (6.4128) | 67.143 (11.4546)
  DAY 1, 24 Hours | 63.400 (7.1992) | 61.267 (7.6295) | 64.071 (11.5190)
  DAY 1, 48 Hours | 64.333 (6.7259) | 63.533 (6.4572) | 63.286 (10.5278)
  DAY 1, 72 Hours | 62.267 (6.9639) | 62.467 (8.0166) | 62.286 (11.0900)

32. Secondary Outcome: Part 1: Change From Baseline in Pulse Rate
Description: Pulse rate was measured in supine position after 10 minutes rest for the participant at indicated time points. Baseline was defined as the latest pre-dose assessment, including those from unscheduled visits. Change from Baseline was defined as any visit value minus Baseline value.
Time Frame: Baseline (Day -1) and 1, 2, 4, 6, 8, 12, 24, 48, 72 Hours on Day 1
Population: Safety Population
Measure: Mean (Standard Deviation); unit: Beats per minute
Arm/Group | Part 1: GSK2838232 200 mg/Ritonavir Capsule Fed | Part 1: GSK2838232 200 mg/Ritonavir Tablet Fed | Part 1: GSK 200 mg/Ritonavir Tablet Fasted
Number analyzed (Participants) | 15 | 15 | 14
Beats per minute
  DAY 1, 1 Hour | 9.644 (9.2897) | 8.023 (9.3536) | -1.286 (4.4390)
  DAY 1, 2 Hours | 7.644 (10.5927) | 8.623 (8.8718) | 0.357 (5.2912)
  DAY 1, 4 Hours | 3.111 (7.1157) | 5.156 (10.5863) | 1.357 (4.6853)
  DAY 1, 6 Hours | 3.844 (8.0953) | 3.823 (11.4959) | 6.643 (2.4580)
  DAY 1, 8 Hours | 1.511 (9.0965) | 2.623 (9.1496) | 3.714 (5.1408)
  DAY 1, 12 Hours | -0.156 (8.6466) | 1.556 (7.3741) | 7.286 (8.0517)
  DAY 1, 24 Hours | -1.623 (8.9894) | -3.044 (8.7852) | 4.214 (6.3150)
  DAY 1, 48 Hours | -0.689 (8.0818) | -0.777 (7.8056) | 3.429 (7.7752)
  DAY 1, 72 Hours | -2.756 (9.7834) | -1.844 (7.4755) | 2.429 (6.6210)

33. Secondary Outcome: Part 1: Number of Participants With Abnormal ECG Findings
Description: Single and triplicate 12-lead ECG's were obtained at least 5 minutes apart in the supine position after 10 minutes of rest at indicated time points using an ECG machine that automatically calculates the heart rate and measures PR, QRS, QT and QTcF intervals. CS and NCS abnormal ECG findings have been presented. CS abnormal findings are those which are not associated with the underlying disease, unless judged by the investigator to be more severe than expected for the participant's condition.
Time Frame: Day -2, Day -1; 1, 2, 4, 6, 8, , 12, 24, 48, 72 hours on Day 1
Population: Safety Population. Only those participants with data available at the specified data points were analyzed (represented by n= X in the category titles).
Measure: Count of Participants; unit: Participants
Arm/Group | Part 1: GSK2838232 200 mg/Ritonavir Capsule Fed | Part 1: GSK2838232 200 mg/Ritonavir Tablet Fed | Part 1: GSK2838232 200 mg/Ritonavir Tablet Fasted
Number analyzed (Participants) | 15 | 15 | 14
Participants
  NCS: DAY -2; n=15, 15, 14 | 10 | 9 | 9
  CS: DAY -2; n=15, 15, 14 | 0 | 0 | 0
  NCS: DAY -1; n=15, 14, 14: number analyzed (Participants) | 15 | 14 | 14
  NCS: DAY -1; n=15, 14, 14 | 7 | 9 | 12
  CS: DAY -1; n=15, 14, 14: number analyzed (Participants) | 15 | 14 | 14
  CS: DAY -1; n=15, 14, 14 | 0 | 0 | 0
  NCS: DAY 1, 1 Hour; n=15, 15, 14 | 6 | 5 | 11
  CS: DAY 1, 1 Hour; n=15, 15, 14 | 0 | 0 | 0
  NCS: DAY 1, 2 Hours; n=15, 15, 13: number analyzed (Participants) | 15 | 15 | 13
  NCS: DAY 1, 2 Hours; n=15, 15, 13 | 5 | 5 | 10
  CS: DAY 1, 2 Hours; n=15, 15, 13: number analyzed (Participants) | 15 | 15 | 13
  CS: DAY 1, 2 Hours; n=15, 15, 13 | 0 | 0 | 0
  NCS: DAY 1, 4 Hours; n=15, 13, 14: number analyzed (Participants) | 15 | 13 | 14
  NCS: DAY 1, 4 Hours; n=15, 13, 14 | 5 | 3 | 13
  CS: DAY 1, 4 Hours; n=15, 13, 14: number analyzed (Participants) | 15 | 13 | 14
  CS: DAY 1, 4 Hours; n=15, 13, 14 | 0 | 0 | 0
  NCS: DAY 1, 6 Hours; n=14, 14, 14: number analyzed (Participants) | 14 | 14 | 14
  NCS: DAY 1, 6 Hours; n=14, 14, 14 | 3 | 3 | 5
  CS: DAY 1, 6 Hours; n=14, 14, 14: number analyzed (Participants) | 14 | 14 | 14
  CS: DAY 1, 6 Hours; n=14, 14, 14 | 0 | 0 | 0
  NCS: DAY 1, 8 Hours; n=15, 15, 14 | 7 | 5 | 8
  CS: DAY 1, 8 Hours; n=15, 15, 14 | 0 | 0 | 0
  NCS: DAY 1, 12 Hours; n=15, 14, 14: number analyzed (Participants) | 15 | 14 | 14
  NCS: DAY 1, 12 Hours; n=15, 14, 14 | 7 | 4 | 9
  CS: DAY 1, 12 Hours; n=15, 14, 14: number analyzed (Participants) | 15 | 14 | 14
  CS: DAY 1, 12 Hours; n=15, 14, 14 | 0 | 0 | 0
  NCS: DAY 1, 24 Hours; n=14, 15, 14: number analyzed (Participants) | 14 | 15 | 14
  NCS: DAY 1, 24 Hours; n=14, 15, 14 | 11 | 10 | 10
  CS: DAY 1, 24 Hours; n=14, 15, 14: number analyzed (Participants) | 14 | 15 | 14
  CS: DAY 1, 24 Hours; n=14, 15, 14 | 0 | 0 | 0
  NCS: DAY 1, 48 Hours; n=15, 15, 14 | 8 | 9 | 11
  CS: DAY 1, 48 Hours; n=15, 15, 14 | 0 | 0 | 0
  NCS: DAY 1, 72 Hours; n=15, 15, 14 | 10 | 8 | 11
  CS: DAY 1, 72 Hours; n=15, 15, 14 | 0 | 0 | 0

34. Secondary Outcome: Part 1: Change From Baseline in Mean Heart Rate Values as ECG Parameter
Description: as for outcome 15
Time Frame: Baseline (Day -1) and 1, 2, 4, 6, 8, 12, 24, 48, 72 hours on Day 1
Population: as for outcome 33
Measure: Mean (Standard Deviation); unit: Beats per minute
Arm/Group | Part 1: GSK2838232 200 mg/Ritonavir Capsule Fed | Part 1: GSK2838232 200 mg/Ritonavir Tablet Fed | Part 1: GSK 200 mg/Ritonavir Tablet Fasted
Number analyzed (Participants) | 15 | 15 | 14
Beats per minute
  DAY 1, 1 Hour; n=15,15,14 | 11.623 (3.5038) | 7.955 (7.1040) | -0.642 (3.6609)
  DAY 1, 2 Hours; n=15,15,13: number analyzed (Participants) | 15 | 15 | 13
  DAY 1, 2 Hours; n=15,15,13 | 10.623 (4.8877) | 8.489 (6.5565) | -1.230 (4.3393)
  DAY 1, 4 Hours; n=15,14,14: number analyzed (Participants) | 15 | 14 | 14
  DAY 1, 4 Hours; n=15,14,14 | 4.156 (3.2562) | 2.500 (7.3292) | 2.144 (4.9148)
  DAY 1, 6 Hours; n=14,14,14: number analyzed (Participants) | 14 | 14 | 14
  DAY 1, 6 Hours; n=14,14,14 | 6.072 (3.0746) | 1.643 (7.5799) | 5.786 (2.6441)
  DAY 1, 8 Hours; n=15,15,14 | 2.223 (4.5377) | 1.489 (7.0631) | 2.929 (4.3034)
  DAY 1, 12 Hours; n=15,15,14 | 4.089 (5.0734) | -0.178 (6.3675) | 6.072 (5.5851)
  DAY 1, 24 Hours; n=15,15,14 | -2.377 (6.3879) | -4.711 (7.0854) | 2.786 (4.2971)
  DAY 1, 48 Hours; n=15,15,14 | 1.023 (7.7608) | -2.378 (6.3181) | 2.358 (6.3093)
  DAY 1, 72 Hours; n=15,15,14 | -0.911 (6.1612) | -3.045 (6.1332) | 2.286 (4.8518)

35. Secondary Outcome: Part 1: Change From Baseline in PR Interval, QRS, QT Interval, and QTcF Interval as ECG Parameters
Description: as for outcome 16
Time Frame: Baseline (Day -1) and 1, 2, 4, 6, 8, 12, 24, 48, 72 hours on Day 1
Population: as for outcome 33
Measure: Mean (Standard Deviation); unit: Milliseconds
Arm/Group | Part 1: GSK2838232 200 mg/Ritonavir Capsule Fed | Part 1: GSK2838232 200 mg/Ritonavir Tablet Fed | Part 1: GSK2838232 200 mg/Ritonavir Tablet Fasted
Number analyzed (Participants) | 15 | 15 | 14
Milliseconds
  PR interval; DAY 1, 1 Hour; n= 15,15,14 | -4.667 (8.7068) | -3.067 (8.0354) | -3.000 (4.1236)
  PR interval; DAY 1, 2 Hours; n=15,15,13: number analyzed (Participants) | 15 | 15 | 13
  PR interval; DAY 1, 2 Hours; n=15,15,13 | -6.001 (7.7330) | -8.000 (11.0362) | -1.846 (6.4305)
  PR interval; DAY 1, 4 Hours; n=15,14,14: number analyzed (Participants) | 15 | 14 | 14
  PR interval; DAY 1, 4 Hours; n=15,14,14 | -7.067 (10.2033) | -5.905 (8.8947) | -2.571 (5.2620)
  PR interval; DAY 1, 6 Hours; n=14,14,14: number analyzed (Participants) | 14 | 14 | 14
  PR interval; DAY 1, 6 Hours; n=14,14,14 | -5.286 (8.1501) | -4.048 (7.9887) | -7.286 (6.3330)
  PR interval; DAY 1, 8 Hours; n=15,15,14 | -2.267 (9.6666) | 0.267 (9.2972) | -7.571 (5.4017)
  PR interval; DAY 1, 12 Hours; n=15,15,14 | 3.599 (7.2967) | 3.600 (10.7074) | -5.143 (5.5061)
  PR interval; DAY 1, 24 Hours; n=15,15,14 | 0.133 (6.2540) | 0.667 (11.6569) | -4.000 (5.2761)
  PR interval; DAY 1, 48 Hours; n=15,15,14 | 0.533 (9.8492) | 0.267 (9.7100) | -2.857 (4.9369)
  PR interval; DAY 1, 72 Hours; n=15,15,14 | 0.266 (6.7270) | -0.800 (8.3925) | 0.286 (9.5887)
  QRS interval; DAY 1, 1 Hour; n=15,15,14 | 0.177 (4.0981) | -1.067 (2.1485) | -1.191 (2.1266)
  QRS interval; DAY 1, 2 Hours; n=15,15,13: number analyzed (Participants) | 15 | 15 | 13
  QRS interval; DAY 1, 2 Hours; n=15,15,13 | -1.289 (2.7414) | -3.601 (5.5916) | -1.949 (3.6451)
  QRS interval; DAY 1, 4 Hours; n=15,14,14: number analyzed (Participants) | 15 | 14 | 14
  QRS interval; DAY 1, 4 Hours; n=15,14,14 | -0.223 (4.7522) | -3.144 (5.5231) | -1.334 (3.5564)
  QRS interval; DAY 1, 6 Hours; n=14,14,14: number analyzed (Participants) | 14 | 14 | 14
  QRS interval; DAY 1, 6 Hours; n=14,14,14 | 1.190 (4.4691) | -1.096 (3.4838) | -0.048 (2.9515)
  QRS interval; DAY 1, 8 Hours; n=15,15,14 | -1.023 (5.4315) | -1.201 (3.2956) | -1.476 (3.0398)
  QRS interval; DAY 1, 12 Hours; n=15,15,14 | 0.577 (5.0503) | 0.266 (3.0628) | -0.905 (2.3614)
  QRS interval; DAY 1, 24 Hours; n=15,15,14 | -0.489 (3.9399) | -0.001 (3.2548) | -1.762 (2.7249)
  QRS interval; DAY 1, 48 Hours; n=15,15,14 | -0.489 (4.0107) | -3.601 (5.2408) | -2.905 (2.8351)
  QRS interval; DAY 1, 72 Hours; n=15,15,14 | 0.311 (3.4718) | -1.067 (4.7049) | -1.905 (2.6381)
  QT interval; DAY 1, 1 Hour; n=15,15,14 | -27.511 (9.5694) | -23.333 (8.8511) | -0.334 (6.8828)
  QT interval; DAY 1, 2 Hours; n=15,15,13: number analyzed (Participants) | 15 | 15 | 13
  QT interval; DAY 1, 2 Hours; n=15,15,13 | -30.844 (12.7773) | -26.266 (8.5061) | 1.435 (9.3833)
  QT interval; DAY 1, 4 Hours; n=15,14,14: number analyzed (Participants) | 15 | 14 | 14
  QT interval; DAY 1, 4 Hours; n=15,14,14 | -17.377 (12.8317) | -15.523 (12.6937) | -2.191 (12.9124)
  QT interval; DAY 1, 6 Hours; n=14,14,14: number analyzed (Participants) | 14 | 14 | 14
  QT interval; DAY 1, 6 Hours; n=14,14,14 | -15.524 (10.6107) | -10.619 (14.9602) | -23.334 (16.4029)
  QT interval; DAY 1, 8 Hours; n=15,15,14 | -9.511 (12.7754) | -6.266 (16.7718) | -12.762 (13.2960)
  QT interval; DAY 1, 12 Hours; n=15,15,14 | -16.044 (19.7270) | -9.466 (15.0727) | -24.334 (22.8434)
  QT interval; DAY 1, 24 Hours; n=15,15,14 | -2.044 (14.0881) | 0.801 (12.2568) | -11.476 (12.3125)
  QT interval; DAY 1, 48 Hours; n=15,15,14 | -3.644 (17.8393) | -0.666 (14.5496) | -7.476 (12.3459)
  QT interval; DAY 1, 72 Hours; n=15,15,14 | -0.977 (15.5657) | 0.134 (13.0685) | -12.762 (15.3517)
  QTcF interval; DAY 1, 1 Hour; n=15,15,14 | -4.666 (10.4724) | -8.868 (7.0866) | -2.285 (11.8494)
  QTcF interval; DAY 1, 2 Hours; n=15,15,13: number analyzed (Participants) | 15 | 15 | 13
  QTcF interval; DAY 1, 2 Hours; n=15,15,13 | -10.133 (10.8407) | -11.068 (8.0958) | -2.076 (12.2719)
  QTcF interval; DAY 1, 4 Hours; n=15,14,14: number analyzed (Participants) | 15 | 14 | 14
  QTcF interval; DAY 1, 4 Hours; n=15,14,14 | -8.466 (10.1552) | -11.335 (10.1802) | 1.858 (10.9901)
  QTcF interval; DAY 1, 6 Hours; n=14,14,14: number analyzed (Participants) | 14 | 14 | 14
  QTcF interval; DAY 1, 6 Hours; n=14,14,14 | -3.714 (9.3976) | -7.573 (12.1949) | -10.499 (12.0696)
  QTcF interval; DAY 1, 8 Hours; n=15,15,14 | -4.333 (11.3261) | -3.268 (14.6848) | -6.356 (11.4959)
  QTcF interval; DAY 1, 12 Hours; n=15,15,14 | -7.199 (11.5629) | -9.735 (15.8796) | -11.214 (12.2055)
  QTcF interval; DAY 1, 24 Hours; n=15,15,14 | -6.933 (10.7150) | -9.601 (9.4605) | -5.856 (9.6316)
  QTcF interval; DAY 1, 48 Hours; n=15,15,14 | -0.999 (12.4826) | -5.601 (5.4868) | -3.785 (9.7479)
  QTcF interval; DAY 1, 72 Hours; n=15,15,14 | -2.466 (9.5081) | -6.401 (10.0613) | -7.785 (12.1949)

36. Secondary Outcome: Part 1: Tlag Following Administration of GSK2838232 Tablet and Capsule Formulation in Fed State and Tablet Formulation in Fasted State
Description: Blood samples were collected at indicated time points for pharmacokinetic analysis of GSK2838232 given as capsule and tablet formulation in fed state as well as tablet formulation in fasted state. Tlag is a time delay between drug administration and first observed concentration. Pharmacokinetic parameters were determined using standard non-compartmental methods.
Time Frame: as for outcome 3
Population: Pharmacokinetic Population
Measure: Median (Full Range); unit: Hours
Arm/Group | Part 1: GSK2838232 200 mg/Ritonavir Capsule Fed | Part 1: GSK2838232 200 mg/Ritonavir Tablet Fed | Part 1: GSK2838232 200 mg/Ritonavir Tablet Fasted
Number analyzed (Participants) | 15 | 15 | 14
Hours | 1.000 [0.00 to 2.00] | 1.000 [0.00 to 3.50] | 0.500 [0.00 to 1.00]

37. Secondary Outcome: Part 1: Tmax Following Administration of GSK2838232 Tablet and Capsule Formulation in Fed State and Tablet Formulation in Fasted State
Description: Blood samples were collected at indicated time points for pharmacokinetic analysis of GSK2838232 given as capsule and tablet formulation in fed state as well as tablet formulation in fasted state. Pharmacokinetic parameters were determined using standard non-compartmental methods.
Time Frame: as for outcome 3
Population: Pharmacokinetic Population
Measure: Median (Full Range); unit: Hours
Arm/Group | Part 1: GSK2838232 200 mg/Ritonavir Capsule Fed | Part 1: GSK2838232 200 mg/Ritonavir Tablet Fed | Part 1: GSK 200 mg/Ritonavir Tablet Fasted
Number analyzed (Participants) | 15 | 15 | 14
Hours | 11.967 [1.50 to 24.02] | 5.983 [2.00 to 24.03] | 3.508 [2.00 to 11.97]

38. Secondary Outcome: Part 1: T1/2 Following Administration of GSK2838232 Tablet and Capsule Formulation in Fed State and Tablet Formulation in Fasted State
Description: as for outcome 37
Time Frame: as for outcome 3
Population: Pharmacokinetic Population
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: Hours
Arm/Group | Part 1: GSK2838232 200 mg/Ritonavir Capsule Fed | Part 1: GSK2838232 200 mg/Ritonavir Tablet Fed | Part 1: GSK 200 mg/Ritonavir Tablet Fasted
Number analyzed (Participants) | 15 | 15 | 14
Hours | 15.606 (14.84) | 15.692 (17.28) | 17.061 (19.01)

39. Secondary Outcome: Part 1: Tlast Following Administration of GSK2838232 Tablet and Capsule Formulation in Fed State and Tablet Formulation in Fasted State
Description: as for outcome 37
Time Frame: as for outcome 3
Population: Pharmacokinetic Population
Measure: Median (Full Range); unit: Hours
Arm/Group | Part 1: GSK2838232 200 mg/Ritonavir Capsule Fed | Part 1: GSK2838232 200 mg/Ritonavir Tablet Fed | Part 1: GSK 200 mg/Ritonavir Tablet Fasted
Number analyzed (Participants) | 15 | 15 | 14
Hours | 119.983 [119.80 to 120.20] | 119.983 [119.70 to 120.08] | 120.017 [95.87 to 120.42]

40. Secondary Outcome: Part 1: Plasma Drug Concentration at 24 Hours (C24) Following Administration of GSK2838232 Tablet and Capsule Formulation in Fed State and Tablet Formulation in Fasted State
Description: as for outcome 37
Time Frame: as for outcome 3
Population: Pharmacokinetic Population
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: Nanograms per milliliter
Arm/Group | Part 1: GSK2838232 200 mg/Ritonavir Capsule Fed | Part 1: GSK2838232 200 mg/Ritonavir Tablet Fed | Part 1: GSK 200 mg/Ritonavir Tablet Fasted
Number analyzed (Participants) | 15 | 15 | 14
Nanograms per milliliter | 84.536 (41.93) | 75.643 (32.57) | 26.852 (35.39)

41. Secondary Outcome: Part 1: AUC(0-t) Following Administration of GSK2838232 Tablet and Capsule Formulation in Fed State and Tablet Formulation in Fasted State
Description: as for outcome 37
Time Frame: as for outcome 3
Population: Pharmacokinetic Population
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: Hours* nanograms per milliliter
Arm/Group | Part 1: GSK2838232 200 mg/Ritonavir Capsule Fed | Part 1: GSK2838232 200 mg/Ritonavir Tablet Fed | Part 1: GSK2838232 200 mg/Ritonavir Tablet Fasted
Number analyzed (Participants) | 15 | 15 | 14
Hours* nanograms per milliliter | 4595.35 (40.28) | 4371.47 (30.03) | 1776.21 (36.60)

42. Secondary Outcome: Part 2: Slope of Pre-dose Concentration of GSK2838232 Administered as Non-boosted Once-daily Doses of a Tablet Formulation to Assess Achievement of Steady State
Description: Blood sample were collected at indicated time points to assess pre-dose concentration of GSK2838232 when administered as non-boosted once-daily doses of a tablet formulation for 11 days in Part 2. Slope and 90 percent confidence interval have been presented.
Time Frame: Pre-dose on Day 3, Day 4, Day 5, Day 6, Day 7, Day 8, Day 9, Day 10 and Day 11 in Part 2
Population: Pharmacokinetic Population
Measure: Number (90% Confidence Interval); unit: Nanograms per milliliter per study day
Arm/Group | Part 2: GSK2838232 500 mg Tablet Fed
Number analyzed (Participants) | 7
Nanograms per milliliter per study day
  Pre-dose, Days 3-11 | -0.00910 [-0.0239 to 0.00574]
  Pre-dose, Days 4-11 | -0.0150 [-0.0337 to 0.00377]
  Pre-dose, Days 5-11 | -0.0379 [-0.0584 to 0.0174]
  Pre-dose, Days 6-11 | -0.0490 [-0.0717 to -0.0263]
  Pre-dose, Days 7-11 | -0.0679 [-0.0971 to -0.0388]
  Pre-dose, Days 8-11 | -0.0672 [-0.111 to -0.0233]
  Pre-dose, Days 9-11 | -0.107 [-0.182 to -0.0322]
  Pre-dose, Days 10-11 | -0.263 [-0.392 to -0.133]

43. Secondary Outcome: Part 2: Accumulation Ratio Calculated From AUC(0-tau) Following Administration of GSK2838232 as Non-boosted Once-daily Doses of a Tablet Formulation
Description: Blood sample were collected at indicated time points to calculate accumulation ratio from AUC(0-tau) following administration of GSK2838232 as non-boosted once-daily doses of a tablet formulation. Accumulation ratio of GSK2838232 was evaluated by Day 11, AUC (0-tau) divided by Day 1, AUC (0-tau).
Time Frame: as for outcome 17
Population: Pharmacokinetic Population
Measure: Mean (Standard Deviation); unit: Ratio of AUC
Arm/Group | Part 2: GSK2838232 500 mg Tablet Fed
Number analyzed (Participants) | 7
Ratio of AUC | 1.3340 (0.18272)

44. Secondary Outcome: Part 2: Accumulation Ratio Calculated From Cmax Following Administration of GSK2838232 as Non-boosted Once-daily Doses of a Tablet Formulation
Description: Blood sample were collected at indicated time points to calculate accumulation ratio from Cmax following administration of GSK2838232 as non-boosted once-daily doses of a tablet formulation. Accumulation ratio of GSK2838232 was evaluated by Day 11, Cmax divided by Day 1, Cmax.
Time Frame: as for outcome 17
Population: Pharmacokinetic Population
Measure: Mean (Standard Deviation); unit: Ratio of Cmax
Arm/Group | Part 2: GSK2838232 500 mg Tablet Fed
Number analyzed (Participants) | 7
Ratio of Cmax | 1.2118 (0.28582)

45. Secondary Outcome: Part 2: Accumulation Ratio Calculated From Ctau Following Administration of GSK2838232 as Non-boosted Once-daily Doses of a Tablet Formulation
Description: Blood sample were collected at indicated time points to calculate accumulation ratio from Ctau following administration of GSK2838232 as non-boosted once-daily doses of a tablet formulation. Accumulation ratio of GSK2838232 was evaluated by Day 11, Ctau divided by Day 1, Ctau.
Time Frame: as for outcome 17
Population: Pharmacokinetic Population
Measure: Mean (Standard Deviation); unit: Ratio of Ctau
Arm/Group | Part 2: GSK2838232 500 mg Tablet Fed
Number analyzed (Participants) | 7
Ratio of Ctau | 1.3205 (0.32907)

ADVERSE EVENTS:
Time Frame: Serious adverse events (SAEs) and Non-SAEs were collected up to 60 days in Part 1 of the study and up to 25 days in Part 2 of the study.
Description: SAEs and Non-SAEs were reported for the Safety Population which comprised of all participants who received at least 1 dose of the study treatment (including placebo) with at least 1 post-Baseline safety assessment.
Arm/Group | Part 1: GSK2838232 200 mg/Ritonavir Capsule Fed | Part 1: GSK2838232 200 mg/Ritonavir Tablet Fed | Part 1: GSK 200 mg/Ritonavir Tablet Fasted | Part 2: Placebo | Part 2: GSK2838232 500 mg Tablet Fed
All-Cause Mortality (participants affected / at risk) | 0/15 | 0/15 | 0/14 | 0/3 | 0/7
Serious Adverse Events (participants affected / at risk) | 0/15 | 0/15 | 0/14 | 0/3 | 0/7
Other Adverse Events (participants affected / at risk) | 3/15 | 2/15 | 1/14 | 1/3 | 0/7
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Part 1: GSK2838232 200 mg/Ritonavir Capsule Fed (N=15) | Part 1: GSK2838232 200 mg/Ritonavir Tablet Fed (N=15) | Part 1: GSK 200 mg/Ritonavir Tablet Fasted (N=14) | Part 2: Placebo (N=3) | Part 2: GSK2838232 500 mg Tablet Fed (N=7)
Abdominal discomfort (Gastrointestinal disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Abdominal pain (Gastrointestinal disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Abdominal pain lower (Gastrointestinal disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Constipation (Gastrointestinal disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Diarrhoea (Gastrointestinal disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Flatulence (Gastrointestinal disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Vomiting (Gastrointestinal disorders) | 1 (2) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Chest discomfort (General disorders) | 0 (0) | 1 (2) | 0 (0) | 0 (0) | 0 (0)
Chills (General disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Infusion site pain (General disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Skin abrasion (Injury, poisoning and procedural complications) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Pain in extremity (Musculoskeletal and connective tissue disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Headache (Nervous system disorders) | 3 (3) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Syncope (Nervous system disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Cough (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
GSK agreements may vary with individual investigators, but will not prohibit any investigator from publishing. GSK supports the publication of results from all centers of a multi-center trial but requests that reports based on single-site data not precede the primary publication of the entire clinical trial.

DOCUMENTS (2):
  • Study Protocol (2017-07-18): https://cdn.clinicaltrials.gov/large-docs/36/NCT03234036/Prot_000.pdf
  • Statistical Analysis Plan (2017-12-07): https://cdn.clinicaltrials.gov/large-docs/36/NCT03234036/SAP_001.pdf